CLINICAL TRIAL: NCT02367781
Title: A Phase III Multicenter, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Atezolizumab (MPDL3280A, Anti-PD-L1 Antibody) in Combination With Carboplatin+Nab-Paclitaxel for Chemotherapy-Naive Patients With Stage IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab in Combination With Carboplatin Plus (+) Nab-Paclitaxel Compared With Carboplatin+Nab-Paclitaxel in Participants With Stage IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Acronym: IMpower130
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29537; 2014-003206-32 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Carcinoma, Non-Squamous Non-Small Cell Lung
MeSH Terms: conditions — Carcinoma | interventions — atezolizumab; Carboplatin; 130-nm albumin-bound paclitaxel; Pemetrexed

ARMS (2):
- Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) (Experimental): Participants received intravenous (IV) infusion of atezolizumab and carboplatin on Day 1 of each 21-day cycle, and nab-paclitaxel on Days 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles or until loss of clinical benefit whichever occurred first during induction treatment phase. Participants received IV infusion of atezolizumab during maintenance treatment phase until loss of clinical benefit.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Carboplatin; Drug: Nab-Paclitaxel
- Arm B (Nab-Paclitaxel+Carboplatin) (Active Comparator): Participants received IV infusion of carboplatin on Day 1 and nab-paclitaxel on Days 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles or until disease progression whichever occurred first during induction treatment phase. Participants received best supportive care during maintenance treatment phase. Switch maintenance to pemetrexed was also permitted. Participants who were consented prior to approval of protocol Version 5 were given the option to cross over to receive atezolizumab as monotherapy until disease progression.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody; Drug: Carboplatin; Drug: Nab-Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab was administered as IV infusion at a dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle. Atezolizumab was administered to participants who were randomized to "Arm A (Atezolizumab + Nab-Paclitaxel + Carboplatin)" and to participants in "Arm B (Nab-Paclitaxel + Carboplatin)" who cross over at progression.
  Other Names: MPDL3280A, RO5541267, Tecentriq
Drug: Carboplatin — Carboplatin was administered at area under the concentration curve (AUC) 6 milligrams per milliliter per minute (mg/mL/min) on Day 1 of each 21-day cycle.
Drug: Nab-Paclitaxel — Nab-paclitaxel was administered as IV infusion at a dose of 100 milligrams per square meter (mg/m^2) on Days 1, 8, and 15 of each 21-day cycle.
Drug: Pemetrexed — Switch maintenance to pemetrexed can be administered within 6 weeks of Day 1 of the last induction cycle.
  Arms: Arm B (Nab-Paclitaxel+Carboplatin)

SUMMARY:
This randomized Phase III, multicenter, open-label study designed to evaluate the safety and efficacy of atezolizumab (an engineered anti-programmed death-ligand 1 [PD-L1] antibody) in combination with carboplatin+nab-paclitaxel compared with treatment with carboplatin+nab-paclitaxel in chemotherapy-naive participants with Stage IV non-squamous NSCLC. Participants were randomized in a 2:1 ratio to Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) or Arm B (Nab-Paclitaxel+Carboplatin).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status of 0 or 1
* Histologically or cytologically confirmed, Stage IV non-squamous NSCLC
* Participants with no prior treatment for Stage IV non-squamous NSCLC
* Previously obtained archival tumor tissue or tissue obtained from fresh biopsy at screening
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function

Exclusion Criteria:

Cancer-Specific Exclusions:

* Active or untreated central nervous system metastases
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome

General Medical Exclusions:

* Pregnant or lactating women
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Severe infection within 4 weeks prior to randomization
* Significant cardiovascular disease
* Illness or condition that interferes with the participant's capacity to understand, follow and/or comply with study procedures

Exclusion Criteria Related to Medications:

* Prior treatment with cluster of differentiation 137 agonists or immune checkpoint blockade therapies, anti-programmed death-1, and anti-PD-L1 therapeutic antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (132):
- United States (57):
  - Highlands Oncology Group, Springdale, Arkansas
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Kaiser Permanente - Sacramento Medical Center and Medical Offices, Sacramento, California
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - Kaiser Permanente - San Jose Medical Center, San Jose, California
  - Kaiser Permanente - San Leandro Medical Center, San Leandro, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Kaiser Permanente - South San Francisco, South San Francisco, California
  - Kaiser Permanente; Oncology Clinical Trials, Vallejo, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Eastern Connecticut Hematology and Oncology Associates; (ECHO), Norwich, Connecticut
  - University of Miami School of Medicine - Sylvester at Deerfield, Deerfield Beach, Florida
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Hospital, Orlando, Florida
  - Florida Cancer Specialists (St. Petersburg - St. Anthony's Professional Building), St. Petersburg, Florida
  - SCRI Florida Cancer Specialists East, West Palm Beach, Florida
  - University Cancer & Blood Center, LLC; Research, Athens, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Carrollton, Georgia
  - Suburban Hematology / Oncology Associates, Lawrenceville, Georgia
  - Southeastern Regional Medical Center, Inc., Newnan, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology; Associates, Ltd., Joliet, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Southern Illinois University, Simmons Cancer Institute, Springfield, Illinois
  - Fort Wayne Med Oncology & Hematology Inc, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Lahey Clinic Med Ctr, Lexington, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Southcoast Health System, Fairhaven, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hematology and Oncology Associates at Bridgepoint, Tupelo, Mississippi
  - Southeast Nebraska Cancer Ctr, Lincoln, Nebraska
  - Va Sierra Nevada Health Care System, Reno, Nevada
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Cancer Inst. of New Jersey, New Brunswick, New Jersey
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Clinical Research Alliance, Westbury, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center; Department of Medicine, Durham, North Carolina
  - W.G. Bill Hefner VA Medical Center, Salisbury, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Mark H. Zangmeister Center, Columbus, Ohio
  - Oncology Hematology Care, Inc., Hamilton, Ohio
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Greenville Health System; Cancer Center, Greenville, South Carolina
  - University Oncology Associates, Chattanooga, Tennessee
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - SCRI The Center For Cancer and Blood Disorders, Denton, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Cancer Care Network of South Texas - SAT & BC, San Antonio, Texas
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - CHU Ambroise Paré, Mons
  - Werken Glorieux VZW, Ronse
  - GasthuisZusters Antwerpen, Wilrijk
- Canada (5):
  - BC Cancer - Surrey, Surrey, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health Centre, Etobicoke, Ontario
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
- France (12):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Institut Hospitalier Franco-Britannique; Cancerologie, Levallois-Perret
  - Fondation Hopital Saint Joseph;Cardiologie Clinique, Marseille
  - Clinique Clementville; Hopital De Jour, Montpellier
  - Centre D'oncologie de Gentilly; Service Oncologie Medicale, Nancy
  - Clinique Catherine de Sienne, Nantes
  - Hopital American de Paris (American Hospital of Paris), Neuilly-sur-Seine
  - HOPITAL DE LA SOURCE; Service de Cardiologie, Point Jaune, Orléans
  - Hopital Pontchaillou, Rennes
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Centre Hospitalier Regional Sud Reunion; Service de Pneumologie, Saint-Pierre
  - CHRU Nancy; Pneumologie, Vandœuvre-lès-Nancy
- Germany (25):
  - Charite - Universitätsmedizin Berlin; Klinik fur Infektiologie und Pneumologie, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Bezirksklinikum Obermain, Ebensfeld
  - Helios Klinikum Erfurt, Erfurt
  - St. Antonius Hospital, Eschweiler
  - Klinikum Esslingen GmbH; Frauenklinik, Esslingen am Neckar
  - Malteser Krankenhaus St. Franziskus-Hospital, Flensburg
  - Krankenhaus Nordwest, Frankfurt am Main
  - Asklepios Fachkliniken GmbH, Gauting
  - SRH Wald-Klinikum Gera; Klinik für Hautkrankheiten und Allergologie, Gera
  - Robert Bosch Krankenhaus; Pneumologie und pneumologische Onkologie, Gerlingen
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - St. Vincentius Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel; Hautklinik, Kassel
  - Katholisches Klinikum Marienhof, Koblenz Am Rhein
  - Universitatsklinikum Schleswig-Holstein; Klinik fuer Innere Medizin I, Lübeck
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - LMU Klinikum der Universitat Munchen, München
  - Universitätsklinikum Tübingen, Tübingen
  - Praxis fur Haematologie und Internistische Onkologie, Velbert
  - Schwarzwald-Baar Klinikum/VS GmbH; Onkologie/Hämatologie/Infektologie, Villingen-Schwenningen
  - Helios Klinik Wuppertal, Wuppertal
- Israel (10):
  - Assaf Harofeh Medical Center, Beer Yaakov
  - Soroka University Medical Centre, Beersheba
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petach Tiqwa
  - Chaim Sheba Medical Center, Ramat Gan
  - Rambam Health Corporation; Oncology Institute, Rambam
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Ctr; Oncology, Tel Aviv
- Italy (6):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino, Campania
  - Azienda Osp Uni Seconda Università Degli Studi Di Napoli; Unità Operativa Oncologia Medica, Napoli, Campania
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - Ospedale Di Macerata; Oncologia, Macerata, The Marches
  - Ospedale Santa Maria Della; Misericordia Di Perugia; Farmacia Ospedaliera, Perugia, Umbria
- Spain (13):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Consorcio Hospitalario Provincial de Castellon, Castellon de LA Plana/castello de LA Plana, Castellon
  - Complejo Hospitalario Universitario A Coruña, A Coruña, LA Coruña
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Hospital Universitario de Canarias, S. Cristobal de La Laguna, Tenerife
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital de San Pedro de Alcantara, Cáceres
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital General Universitario de Valencia, Valencia
  - Hospital NisA 9 de Octubre, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza

REFERENCES:
- [Derived] Socinski MA, Jotte RM, Cappuzzo F, Nishio M, Mok TSK, Reck M, Finley GG, Kaul MD, Yu W, Paranthaman N, Bara I, West HJ. Association of Immune-Related Adverse Events With Efficacy of Atezolizumab in Patients With Non-Small Cell Lung Cancer: Pooled Analyses of the Phase 3 IMpower130, IMpower132, and IMpower150 Randomized Clinical Trials. JAMA Oncol. 2023 Apr 1;9(4):527-535. doi: 10.1001/jamaoncol.2022.7711. PMID 36795388
- [Derived] Ton TGN, Pal N, Trinh H, Mahrus S, Bretscher MT, Machado RJM, Sadetsky N, Chaudhary N, Lu MW, Riely GJ. Replication of Overall Survival, Progression-Free Survival, and Overall Response in Chemotherapy Arms of Non-Small Cell Lung Cancer Trials Using Real-World Data. Clin Cancer Res. 2022 Jul 1;28(13):2844-2853. doi: 10.1158/1078-0432.CCR-22-0471. PMID 35511917
- [Derived] West H, McCleod M, Hussein M, Morabito A, Rittmeyer A, Conter HJ, Kopp HG, Daniel D, McCune S, Mekhail T, Zer A, Reinmuth N, Sadiq A, Sandler A, Lin W, Ochi Lohmann T, Archer V, Wang L, Kowanetz M, Cappuzzo F. Atezolizumab in combination with carboplatin plus nab-paclitaxel chemotherapy compared with chemotherapy alone as first-line treatment for metastatic non-squamous non-small-cell lung cancer (IMpower130): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Jul;20(7):924-937. doi: 10.1016/S1470-2045(19)30167-6. Epub 2019 May 20. PMID 31122901

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in this study included: histologically or cytologically confirmed, Stage IV non-squamous NSCLC; and no prior treatment for Stage IV non-squamous NSCLC.
  At the time of study completion a few participants that were still on maintenance treatment with atezolizumab were moved to another study, Post-Trial Access Program, or commercial use. Therefore, the reason for discontinuation was entered "Study terminated by Sponsor" for these participants.
Groups:
- Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin): Participants received intravenous (IV) infusion of atezolizumab and carboplatin on Day 1 of each 21-day cycle, and nab-paclitaxel on Days 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles or until loss of clinical benefit whichever occurs first during induction treatment phase. Participants received IV infusion of atezolizumab during maintenance treatment phase until loss of clinical benefit.
- Arm B (Nab-Paclitaxel+Carboplatin): Participants received IV infusion of carboplatin on Day 1 and nab-paclitaxel on Days 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles or until disease progression whichever occurs first during induction treatment phase. Participants will receive best supportive care during maintenance treatment phase. Switch maintenance to pemetrexed is also permitted. Participants who were consented prior to approval of protocol Version 5 will be given the option to cross over to receive atezolizumab as monotherapy until disease progression.
Period: Overall Study
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Started | 483 | 240
Completed | 0 | 0
Not Completed | 483 | 240
Not completed — Withdrawal by Subject | 20 | 13
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 7 | 0
Not completed — Randomized in Error | 5 | 4
Not completed — Non-Compliance | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 330 | 176
Not completed — Patient Moving to Roll-Over Study | 17 | 5
Not completed — Prolonged Hospitalization | 1 | 0
Not completed — Death Prior First Dose | 1 | 0
Not completed — Administrative-Change Facility | 1 | 0
Not completed — Request From Sponsor to Withdraw Patient in Survival Follow-Up | 78 | 29
Not completed — Patient Moved to Commercial Atezolizumab Use | 14 | 9
Not completed — Study Terminated by Sponsor | 3 | 1
Not completed — Patient Admitted to Hospital & Couldn't be Dosed for Randomization | 1 | 0
Not completed — Sponsor Decision | 2 | 0
Not completed — 3 Year Treatment Completed, Immunotherapy Paused, Continuing Follow-Up Planned | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin) | Total
Number analyzed (Participants) | 483 | 240 | 723
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (9.5) | 64.4 (8.9) | 64.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 102 | 308
  Male | 277 | 138 | 415
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 12 | 37
  Not Hispanic or Latino | 426 | 213 | 639
  Unknown or Not Reported | 32 | 15 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 8 | 26
  White | 428 | 222 | 650
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 21 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in the ITT-WT Population
Description: PFS is defined as the time between the date of randomization and the date of first documented disease progression as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurs first in the ITT-WT population.
Time Frame: Up to approximately 35 months after first patient enrolled
Population: The ITT- WT population was defined as the ITT population excluding participants with an activating EGFR mutation or ALK translocation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 456 | 229
Months | 7.0 [6.3 to 7.3] | 5.5 [4.4 to 5.9]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.639, 95% CI 2-sided [0.536 to 0.763]

2. Primary Outcome: Overall Survival (OS) in the ITT-WT Population
Description: OS is defined as the time between the date of randomization and date of death from any cause in the ITT-WT population.
Time Frame: Up to approximately 35 months after first patient enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 456 | 229
Months | 18.6 [15.8 to 21.2] | 13.9 [12.0 to 18.7]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Test type: Superiority — Stratified Analysis; p = 0.0298, Log Rank; Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.636 to 0.977]

3. Secondary Outcome: PFS as Determined by the Investigator Using Recist v1.1 in the ITT Population, PD-L1 Expression Population, and PD-L1 Expression WT Population
Description: PFS is defined as the time between the date of randomization and the date of first documented disease progression as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurs first. The ITT population was defined as all randomized participants, regardless of receipt of the assigned treatment. The PD-L1 expression population is defined as one of the following: PD-L1 IHC TC1/2/3 or IC1/2/3 population, defined as ITT participants with PD-L1 IHC TC1/2/3 or IC1/2/3 expression in baseline tumor tissue; PD-L1 IHC TC2/3 or IC2/3 population, defined as ITT participants with PD-L1 IHC TC2/3 or IC2/3 expression in baseline tumor tissue; PD-L1 IHC TC3 or IC3 population, defined as ITT participants with PD-L1 IHC TC3 or IC3 expression in baseline tumor tissue. The PD-L1 expression WT population is defined as the PD-L1 expression population excluding participants with an activating EGFR mutation or ALK translocation.
Time Frame: Up to approximately 35 months after first subject enrolled
Population: ITT Population, PD-L1 Expression Population, and PD-L1 Expression WT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 483 | 240
Months
  ITT Population | 7.0 [6.3 to 7.3] | 5.6 [4.5 to 5.9]
  TC1/2/3 or IC1/2/3 ITT Population: number analyzed (Participants) | 230 | 111
  TC1/2/3 or IC1/2/3 ITT Population | 7.5 [7.0 to 9.1] | 5.7 [4.5 to 6.6]
  TC1/2/3 or IC1/2/3-WT ITT Population: number analyzed (Participants) | 216 | 107
  TC1/2/3 or IC1/2/3-WT ITT Population | 7.5 [7.0 to 9.0] | 5.9 [4.5 to 6.6]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); ITT Population; Test type: Superiority — Stratified Analysis; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.647, 95% CI 2-sided [0.545 to 0.768]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3-WT ITT Population; Test type: Superiority — Unstratified Analysis; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.561, 95% CI 2-sided [0.432 to 0.728]
Statistical Analysis 3: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 ITT Population; Test type: Superiority — Unstratified Analysis; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.549, 95% CI 2-sided [0.425 to 0.708]

4. Secondary Outcome: OS as Determined by the Investigator Using Recist v1.1 in the ITT Population
Description: OS is defined as the time between the date of randomization and date of death from any cause in the ITT population.
Time Frame: Up to approximately 41 months after first subject enrolled
Population: The ITT population was defined as all randomized participants, regardless of receipt of the assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 483 | 240
Months | 17.0 [14.9 to 19.7] | 13.5 [11.9 to 17.7]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Test type: Superiority — Stratified Analysis; p = 0.0732, Log Rank; Hazard Ratio (HR) = 0.837, 95% CI 2-sided [0.689 to 1.017]

5. Secondary Outcome: OS as Determined by the Investigator Using RECIST v1.1 in the PD-L1 Expression Population and PD-L1 Expression WT Population
Description: OS is defined as the time between the date of randomization and date of death from any cause in the PD-L1 Expression Population and PD-L1 Expression WT Population. The PD-L1 expression population is defined as one of the following: PD-L1 IHC TC1/2/3 or IC1/2/3 population, defined as ITT participants with PD-L1 IHC TC1/2/3 or IC1/2/3 expression in baseline tumor tissue; PD-L1 IHC TC2/3 or IC2/3 population, defined as ITT participants with PD-L1 IHC TC2/3 or IC2/3 expression in baseline tumor tissue; PD-L1 IHC TC3 or IC3 population, defined as ITT participants with PD-L1 IHC TC3 or IC3 expression in baseline tumor tissue. The PD-L1 expression WT population is defined as the PD-L1 expression population excluding participants with an activating EGFR mutation or ALK translocation.
Time Frame: Up to approximately 35 months after first patient enrolled
Population: PD-L1 Expression Population and PD-L1 Expression WT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 230 | 111
Months
  TC1/2/3 or IC1/2/3 ITT Population | 21.2 [17.3 to 28.2] | 16.9 [12.5 to 22.0]
  TC1/2/3 or IC1/2/3 WT ITT Population: number analyzed (Participants) | 216 | 107
  TC1/2/3 or IC1/2/3 WT ITT Population | 21.2 [18.1 to 28.2] | 16.9 [12.5 to 22.0]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 ITT Population; Test type: Superiority — Unstratified Analysis; p = 0.0830, Log Rank; Hazard Ratio (HR) = 0.752, 95% CI 2-sided [0.545 to 1.039]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 WT ITT Population; Test type: Superiority — Unstratified Analysis; p = 0.0813, Log Rank; Hazard Ratio (HR) = 0.746, 95% CI 2-sided [0.536 to 1.038]

6. Secondary Outcome: Percentage of Participants With an Objective Response (OR) (Complete Response [CR] or Partial Response [PR]) as Determined by the Investigator Using RECIST v1.1 in the ITT-WT Population
Description: ORR (confirmation not required) is defined as the proportion of participants with an objective response, either CR or PR, with the use of RECIST v1.1, as determined by the investigator in the ITT-WT population.
Time Frame: Up to approximately 41 months after first subject enrolled
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 452 | 227
Percentage of participants | 60.2 | 41.0
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Test type: Superiority — Stratified Analysis; p < .0001, Cochran-Mantel-Haenszel; Difference in Response Rate = 19.21, 95% CI 2-sided [11.05 to 27.37] — Wald with Continuity Correction

7. Secondary Outcome: Percentage of Participants With an Objective Response (OR) (Complete Response [CR] or Partial Response [PR]) as Determined by the Investigator Using RECIST v1.1 in the ITT Population, PD-L1 Expression Population, and PD-L1 Expression WT Population
Description: ORR (confirmation not required) is defined as proportion of participants with an objective response, either CR or PR, with the use of RECIST v1.1, as determined by investigator in ITT population, PD-L1 Expression population, and PD-L1 Expression WT population. ITT population was defined as all randomized participants, regardless of receipt of the assigned treatment. PD-L1 expression population is defined as one of the following: PD-L1 IHC TC1/2/3 or IC1/2/3 population, defined as ITT participants with PD-L1 IHC TC1/2/3 or IC1/2/3 expression in baseline tumor tissue; PD-L1 IHC TC2/3 or IC2/3 population, defined as ITT participants with PD-L1 IHC TC2/3 or IC2/3 expression in baseline tumor tissue; PD-L1 IHC TC3 or IC3 population, defined as ITT participants with PD-L1 IHC TC3 or IC3 expression in baseline tumor tissue. PD-L1 expression WT population is defined as PD-L1 expression population excluding participants with an activating EGFR mutation or ALK translocation.
Time Frame: Up to approximately 35 months after first subject enrolled
Population: ITT Population, PD-L1 Expression Population, and PD-L1 Expression WT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 479 | 237
Percentage of participants
  ITT Population | 59.1 | 42.2
  TC1/2/3 or IC1/2/3 ITT WT Population: number analyzed (Participants) | 215 | 106
  TC1/2/3 or IC1/2/3 ITT WT Population | 65.6 | 46.2
  TC1/2/3 or IC1/2/3 ITT Population: number analyzed (Participants) | 229 | 109
  TC1/2/3 or IC1/2/3 ITT Population | 64.6 | 45.0
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); ITT Population; Test type: Superiority — Unstratified Analysis; p < .0001, Cochran-Mantel-Haenszel; Difference in Response Rate = 16.89, 95% CI 2-sided [8.90 to 24.88] — Wald with Continuity Correction
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 ITT WT Population; Test type: Superiority — Stratified Analysis; Odds Ratio (OR) = 2.22, 95% CI 2-sided [1.38 to 3.56]
Statistical Analysis 3: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 ITT Population; Test type: Superiority — Stratified Analysis; p = 0.0007, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.39 to 3.51]

8. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator Using RECIST v1.1 in ITT-WT Population, ITT Population, and PD-L1 Expression Population and PD-L1 Expression WT Population
Description: DOR,defined for participants with objective response (OR) as time from 1st documented OR to documented disease progression as determined by investigator using RECIST v1.1,or death from any cause,whichever occurs 1st.ITT defined as all randomized participants,regardless of receipt of assigned treatment.ITT-WT defined as ITT population excluding participants with activating EGFR mutation or ALK translocation.PD-L1 expression population is defined as one of following:PD-L1 IHC TC1/2/3 or IC1/2/3 population,defined as ITT participants with PD-L1 IHC TC1/2/3 or IC1/2/3 expression in baseline tumor tissue;PD-L1 IHC TC2/3 or IC2/3 population, defined as ITT participants with PD-L1 IHC TC2/3 or IC2/3 expression in baseline tumor tissue;PD-L1 IHC TC3 or IC3 population,defined as ITT participants with PD-L1 IHC TC3 or IC3 expression in baseline tumor tissue.PD-L1 expression WT is defined as PD-L1 expression population excluding participants with activating EGFR mutation or ALK translocation.
Time Frame: Up to approximately 35 months after first subject enrolled
Population: ITT-WT Population, ITT Population, and PD-L1 Expression Population and PD-l1 Expression WT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 283 | 100
Months
  ITT Population | 6.2 [5.6 to 7.9] | 5.4 [4.1 to 5.8]
  ITT-WT Population: number analyzed (Participants) | 267 | 93
  ITT-WT Population | 6.7 [5.6 to 8.0] | 5.4 [3.9 to 5.8]
  TC1/2/3 or IC1/2/3 ITT Population: number analyzed (Participants) | 148 | 49
  TC1/2/3 or IC1/2/3 ITT Population | 7.2 [5.7 to 9.0] | 5.0 [3.2 to 6.1]
  TC1/2/3 or IC1/2/3 ITT WT Population: number analyzed (Participants) | 141 | 49
  TC1/2/3 or IC1/2/3 ITT WT Population | 7.2 [5.7 to 9.0] | 5.0 [3.2 to 6.1]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); ITT Population; Test type: Superiority — Unstratified Analysis; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.614, 95% CI 2-sided [0.473 to 0.797]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); ITT-WT Population; Test type: Superiority — Unstratified Analysis; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.600, 95% CI 2-sided [0.458 to 0.785]
Statistical Analysis 3: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 ITT Population; Test type: Superiority — Unstratified Analysis; p = 0.0011, Log Rank; Hazard Ratio (HR) = 0.548, 95% CI 2-sided [0.379 to 0.791]
Statistical Analysis 4: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); TC1/2/3 or IC1/2/3 ITT WT Population; Test type: Superiority — Unstratified Analysis; p = 0.0014, Log Rank; Hazard Ratio (HR) = 0.551, 95% CI 2-sided [0.381 to 0.798]

9. Secondary Outcome: Event Free Rate (%) at Year 1 and 2 in ITT-WT Population and ITT Population
Description: The OS rate at the 1- and 2-year landmark time points after randomization.
Time Frame: Up to 41 months after first patient enrolled, years 1 and 2 reported
Population: The ITT- WT population was defined as the ITT population excluding participants with an activating EGFR mutation or ALK translocation. The ITT population was defined as all randomized participants, regardless of receipt of the assigned treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 483 | 240
Percentage of participants
  Event Free Rate (%) at Year 1 ITT WT: number analyzed (Participants) | 456 | 229
  Event Free Rate (%) at Year 1 ITT WT | 62.02 [57.53 to 66.51] | 54.56 [48.04 to 61.08]
  Event Free Rate (%) at Year 2 ITT WT: number analyzed (Participants) | 456 | 229
  Event Free Rate (%) at Year 2 ITT WT | 40.43 [35.64 to 45.22] | 32.36 [25.80 to 38.92]
  Event Free Rate (%) at Year 1 ITT | 61.65 [57.29 to 66.02] | 54.47 [48.09 to 60.84]
  Event Free Rate (%) at Year 2 ITT | 39.73 [35.10 to 44.37] | 32.21 [25.79 to 38.63]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) at Year 1 ITT WT Population; Test type: Superiority; p = 0.0647, Z-test; Difference in Event Free Rate = 7.46, 95% CI 2-sided [-0.45 to 15.37]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) at Year 2 ITT WT Population; Test type: Superiority; p = 0.0516, Z-test; Difference in Event Free Rate = 8.07, 95% CI 2-sided [-0.06 to 16.19]
Statistical Analysis 3: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) at Year 1 ITT Population; Test type: Superiority; p = 0.0683, Z-test; Difference in Event Free Rate = 7.19, 95% CI 2-sided [-0.54 to 14.91]
Statistical Analysis 4: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) at Year 2 ITT Population; Test type: Superiority; p = 0.0625, Z-test; Difference in Event Free Rate = 7.53, 95% CI 2-sided [-0.39 to 15.44]

10. Secondary Outcome: Event Free Rate (%) at Year 1 and 2 in PD-L1 Expression Population and PD-L1 Expression WT Population
Description: The OS rate at the 1- and 2-year landmark time points after randomization in the PD-L1 Expression Population and PD-L1 Expression WT Population. The PD-L1 expression population is defined as one of the following: PD-L1 IHC TC1/2/3 or IC1/2/3 population, defined as ITT participants with PD-L1 IHC TC1/2/3 or IC1/2/3 expression in baseline tumor tissue; PD-L1 IHC TC2/3 or IC2/3 population, defined as ITT participants with PD-L1 IHC TC2/3 or IC2/3 expression in baseline tumor tissue; PD-L1 IHC TC3 or IC3 population, defined as ITT participants with PD-L1 IHC TC3 or IC3 expression in baseline tumor tissue. The PD-L1 expression WT population is defined as the PD-L1 expression population excluding participants with an activating EGFR mutation or ALK translocation.
Time Frame: Up to 35 months after first patient enrolled, years 1 and 2 reported
Population: PD-L1 Expression Population and PD-L1 Expression WT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 230 | 111
Percentage of participants
  Event Free Rate (%) at Year 1 TC1/2/3 or IC1/2/3 ITT | 68.56 [62.46 to 74.66] | 61.86 [52.55 to 71.17]
  Event Free Rate (%) at Year 2 TC1/2/3 or IC1/2/3 ITT | 44.63 [35.99 to 53.27] | 35.98 [23.25 to 48.72]
  Event Free Rate (%) at Year 1 TC1/2/3 or IC1/2/3 ITT WT: number analyzed (Participants) | 216 | 107
  Event Free Rate (%) at Year 1 TC1/2/3 or IC1/2/3 ITT WT | 68.84 [62.56 to 75.13] | 62.51 [53.07 to 71.94]
  Event Free Rate (%) at Year 2 TC1/2/3 or IC1/2/3 ITT WT: number analyzed (Participants) | 216 | 107
  Event Free Rate (%) at Year 2 TC1/2/3 or IC1/2/3 ITT WT | 44.02 [34.86 to 53.18] | 35.33 [22.06 to 48.60]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) at Year 1 TC1/2/3 or IC1/2/3 ITT; Test type: Superiority; p = 0.2385, Z-test; Difference in Event Free Rate = 6.69, 95% CI 2-sided [-4.44 to 17.83]
Statistical Analysis 2: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) at Year 2 TC1/2/3 or IC1/2/3 ITT; Test type: Superiority; p = 0.2710, Z-test; Difference in Event Free Rate = 8.64, 95% CI 2-sided [-6.75 to 24.03]
Statistical Analysis 3: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) Year 1 TC1/2/3 or IC1/2/3 ITT WT; Test type: Superiority; p = 0.2733, Z-test; Difference in Event Free Rate = 6.34, 95% CI 2-sided [-5.00 to 17.67]
Statistical Analysis 4: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Event Free Rate (%) Year 2 TC1/2/3 or IC1/2/3 ITT WT; Test type: Superiority; p = 0.2909, Z-test; Difference in Event Free Rate = 8.69, 95% CI 2-sided [-7.44 to 24.81]

11. Secondary Outcome: Time to Deterioration (TTD) in Patient-Reported Lung Cancer Symptoms in the ITT-WT Population
Description: Defined as time from randomization to confirmed deterioration (10-point change) on the combined European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core (EORTC QLQ-C30) and supplemental lung cancer module (EORTC QLQ-LC13) symptom subscales.
Time Frame: Up to approximately 35 months after first subject enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 451 | 228
Months | 2.2 [1.8 to 3.1] | 1.9 [1.5 to 2.4]
Statistical Analysis 1: Comparison: Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) vs Arm B (Nab-Paclitaxel+Carboplatin); Test type: Superiority — Stratified Analysis; p = 0.3342, Log Rank; Hazard Ratio (HR) = 0.893, 95% CI 2-sided [0.711 to 1.123]

12. Secondary Outcome: Change From Baseline in Patient-Reported Lung Cancer Symptoms Score Using the Symptoms in Lung Cancer (SILC) Scale
Description: Change from baseline per SILC scale will be analyzed for each lung cancer symptoms scores. SILC questionnaire comprises 3 individual symptoms & are scored at individual symptom level, thus have a dyspnea score, chest pain score, & cough score. There are a total of 9 questions in SILC questionnaire, each question has a minimum value of 0 & maximum value of 4. Each individual symptom score is calculated as average of responses for symptom items. 'Chest pain' score is mean of question 1 & 2, 'Cough' score is mean of question 3 & 4 and 'Dyspnea' score is mean of question 5 to 9 in SILC questionnaire. An increase in score is suggestive of a worsening in symptomology. A score change of ≥0.3 points for dyspnea & cough symptom scores is considered to be clinically significant; whereas a score change of≥0.5 points for chest pain score is considered to be clinically significant.
Time Frame: Up to approximately 35 months after first subject enrolled
Population: Patient-reported outcome (PRO) analysis were conducted on either the ITT-WT population or the PRO-evaluable WT population, defined as participants randomized into the ITT-WT population who completed a given PRO questionnaire at the baseline visit and at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 236 | 129
Units on a scale
  Chest Pain, Week 1: number analyzed (Participants) | 203 | 114
  Chest Pain, Week 1 | 0.19 (0.86) | 0.14 (0.90)
  Chest Pain, Week 2: number analyzed (Participants) | 204 | 108
  Chest Pain, Week 2 | -0.02 (0.89) | 0.03 (0.91)
  Chest Pain, Week 3: number analyzed (Participants) | 197 | 106
  Chest Pain, Week 3 | -0.05 (0.95) | 0.01 (0.92)
  Chest Pain, Week 4: number analyzed (Participants) | 190 | 102
  Chest Pain, Week 4 | -0.11 (0.95) | 0.01 (1.02)
  Chest Pain, Week 5: number analyzed (Participants) | 192 | 97
  Chest Pain, Week 5 | -0.12 (0.99) | 0.00 (1.03)
  Chest Pain, Week 6: number analyzed (Participants) | 182 | 98
  Chest Pain, Week 6 | -0.24 (1.07) | 0.03 (1.03)
  Chest Pain, Week 7: number analyzed (Participants) | 176 | 87
  Chest Pain, Week 7 | -0.23 (1.11) | 0.03 (1.08)
  Chest Pain, Week 8: number analyzed (Participants) | 169 | 80
  Chest Pain, Week 8 | -0.21 (0.99) | -0.14 (1.00)
  Chest Pain, Week 9: number analyzed (Participants) | 172 | 80
  Chest Pain, Week 9 | -0.18 (1.07) | -0.01 (1.07)
  Chest Pain, Week 10: number analyzed (Participants) | 166 | 75
  Chest Pain, Week 10 | -0.10 (1.07) | -0.07 (1.01)
  Chest Pain, Week 11: number analyzed (Participants) | 171 | 78
  Chest Pain, Week 11 | -0.11 (1.14) | 0.01 (0.96)
  Chest Pain, Week 12: number analyzed (Participants) | 160 | 72
  Chest Pain, Week 12 | -0.15 (1.09) | -0.10 (1.13)
  Chest Pain, Week 13: number analyzed (Participants) | 151 | 61
  Chest Pain, Week 13 | -0.26 (1.07) | -0.03 (1.02)
  Chest Pain, Week 14: number analyzed (Participants) | 144 | 62
  Chest Pain, Week 14 | -0.28 (1.08) | -0.17 (1.18)
  Chest Pain, Week 15: number analyzed (Participants) | 143 | 51
  Chest Pain, Week 15 | -0.26 (1.14) | -0.19 (1.19)
  Chest Pain, Week 16: number analyzed (Participants) | 139 | 52
  Chest Pain, Week 16 | -0.33 (1.11) | -0.16 (1.20)
  Chest Pain, Week 17: number analyzed (Participants) | 145 | 53
  Chest Pain, Week 17 | -0.33 (1.11) | -0.14 (1.13)
  Chest Pain, Week 18: number analyzed (Participants) | 136 | 49
  Chest Pain, Week 18 | -0.28 (1.08) | -0.07 (1.13)
  Chest Pain, Week 19: number analyzed (Participants) | 124 | 45
  Chest Pain, Week 19 | -0.28 (1.04) | -0.16 (1.00)
  Chest Pain, Week 20: number analyzed (Participants) | 123 | 43
  Chest Pain, Week 20 | -0.26 (1.03) | -0.22 (1.02)
  Chest Pain, Week 21: number analyzed (Participants) | 126 | 41
  Chest Pain, Week 21 | -0.25 (1.04) | -0.32 (1.08)
  Chest Pain, Week 22: number analyzed (Participants) | 116 | 37
  Chest Pain, Week 22 | -0.28 (1.01) | -0.11 (1.03)
  Chest Pain, Week 23: number analyzed (Participants) | 122 | 35
  Chest Pain, Week 23 | -0.24 (1.03) | -0.19 (1.04)
  Chest Pain, Week 24: number analyzed (Participants) | 110 | 34
  Chest Pain, Week 24 | -0.21 (1.01) | -0.43 (1.03)
  Chest Pain, Week 25: number analyzed (Participants) | 104 | 31
  Chest Pain, Week 25 | -0.20 (0.98) | -0.24 (1.07)
  Chest Pain, Week 26: number analyzed (Participants) | 109 | 31
  Chest Pain, Week 26 | -0.17 (1.01) | -0.13 (0.91)
  Chest Pain, Week 27: number analyzed (Participants) | 102 | 27
  Chest Pain, Week 27 | -0.22 (1.01) | -0.15 (1.17)
  Chest Pain, Week 28: number analyzed (Participants) | 96 | 28
  Chest Pain, Week 28 | -0.20 (0.98) | -0.07 (0.91)
  Chest Pain, Week 29: number analyzed (Participants) | 104 | 27
  Chest Pain, Week 29 | -0.27 (1.09) | -0.04 (0.92)
  Chest Pain, Week 30: number analyzed (Participants) | 100 | 23
  Chest Pain, Week 30 | -0.15 (1.06) | -0.28 (1.12)
  Chest Pain, Week 31: number analyzed (Participants) | 93 | 25
  Chest Pain, Week 31 | -0.16 (0.95) | -0.12 (1.05)
  Chest Pain, Week 32: number analyzed (Participants) | 88 | 25
  Chest Pain, Week 32 | -0.19 (0.89) | -0.30 (1.10)
  Chest Pain, Week 33: number analyzed (Participants) | 88 | 25
  Chest Pain, Week 33 | -0.18 (1.00) | -0.18 (1.11)
  Chest Pain, Week 34: number analyzed (Participants) | 85 | 24
  Chest Pain, Week 34 | -0.18 (1.07) | -0.17 (1.18)
  Chest Pain, Week 35: number analyzed (Participants) | 87 | 20
  Chest Pain, Week 35 | -0.10 (1.09) | 0.05 (1.06)
  Chest Pain, Week 36: number analyzed (Participants) | 85 | 20
  Chest Pain, Week 36 | -0.21 (1.08) | -0.35 (1.01)
  Chest Pain, Week 37: number analyzed (Participants) | 82 | 21
  Chest Pain, Week 37 | -0.18 (1.18) | -0.10 (1.04)
  Chest Pain, Week 38: number analyzed (Participants) | 83 | 19
  Chest Pain, Week 38 | -0.32 (1.02) | -0.05 (1.01)
  Chest Pain, Week 39: number analyzed (Participants) | 78 | 18
  Chest Pain, Week 39 | -0.28 (0.90) | -0.22 (1.06)
  Chest Pain, Week 40: number analyzed (Participants) | 76 | 14
  Chest Pain, Week 40 | -0.19 (0.87) | -0.39 (0.81)
  Chest Pain, Week 41: number analyzed (Participants) | 77 | 16
  Chest Pain, Week 41 | -0.25 (0.93) | -0.19 (0.89)
  Chest Pain, Week 42: number analyzed (Participants) | 70 | 16
  Chest Pain, Week 42 | -0.16 (1.02) | -0.41 (0.74)
  Chest Pain, Week 43: number analyzed (Participants) | 68 | 16
  Chest Pain, Week 43 | -0.24 (0.90) | -0.22 (0.95)
  Chest Pain, Week 44: number analyzed (Participants) | 76 | 16
  Chest Pain, Week 44 | -0.24 (0.95) | 0.00 (0.98)
  Chest Pain, Week 45: number analyzed (Participants) | 69 | 14
  Chest Pain, Week 45 | -0.14 (0.95) | -0.07 (0.78)
  Chest Pain, Week 46: number analyzed (Participants) | 71 | 15
  Chest Pain, Week 46 | -0.15 (0.94) | -0.07 (1.03)
  Chest Pain, Week 47: number analyzed (Participants) | 70 | 13
  Chest Pain, Week 47 | -0.22 (0.98) | -0.15 (0.90)
  Chest Pain, Week 48: number analyzed (Participants) | 66 | 11
  Chest Pain, Week 48 | -0.14 (0.91) | -0.18 (0.98)
  Chest Pain, Week 49: number analyzed (Participants) | 65 | 9
  Chest Pain, Week 49 | -0.22 (0.91) | -0.72 (0.75)
  Chest Pain, Week 50: number analyzed (Participants) | 70 | 8
  Chest Pain, Week 50 | -0.18 (0.91) | -0.19 (0.70)
  Chest Pain, Week 51: number analyzed (Participants) | 65 | 10
  Chest Pain, Week 51 | -0.13 (0.71) | -0.50 (0.78)
  Chest Pain, Week 52: number analyzed (Participants) | 72 | 7
  Chest Pain, Week 52 | -0.15 (0.83) | -0.36 (0.63)
  Chest Pain, Week 53: number analyzed (Participants) | 64 | 6
  Chest Pain, Week 53 | -0.20 (0.82) | -0.33 (0.61)
  Chest Pain, Week 54: number analyzed (Participants) | 65 | 7
  Chest Pain, Week 54 | -0.22 (0.87) | -0.21 (0.70)
  Chest Pain, Week 55: number analyzed (Participants) | 62 | 5
  Chest Pain, Week 55 | -0.34 (0.80) | -0.30 (0.76)
  Chest Pain, Week 56: number analyzed (Participants) | 62 | 6
  Chest Pain, Week 56 | -0.19 (0.95) | -0.33 (0.68)
  Chest Pain, Week 57: number analyzed (Participants) | 62 | 5
  Chest Pain, Week 57 | -0.19 (0.76) | -0.40 (0.65)
  Chest Pain, Week 58: number analyzed (Participants) | 56 | 4
  Chest Pain, Week 58 | -0.32 (0.92) | -0.50 (1.15)
  Chest Pain, Week 59: number analyzed (Participants) | 52 | 4
  Chest Pain, Week 59 | -0.25 (0.93) | -0.63 (0.75)
  Chest Pain, Week 60: number analyzed (Participants) | 48 | 4
  Chest Pain, Week 60 | -0.27 (1.03) | -0.50 (1.08)
  Chest Pain, Week 61: number analyzed (Participants) | 49 | 5
  Chest Pain, Week 61 | -0.28 (1.02) | -0.20 (1.15)
  Chest Pain, Week 62: number analyzed (Participants) | 41 | 5
  Chest Pain, Week 62 | -0.16 (1.06) | -0.40 (1.47)
  Chest Pain, Week 63: number analyzed (Participants) | 43 | 5
  Chest Pain, Week 63 | -0.12 (0.82) | -0.10 (1.34)
  Chest Pain, Week 64: number analyzed (Participants) | 42 | 4
  Chest Pain, Week 64 | -0.15 (0.83) | 0.38 (1.44)
  Chest Pain, Week 65: number analyzed (Participants) | 40 | 3
  Chest Pain, Week 65 | -0.31 (0.84) | 0.17 (1.76)
  Chest Pain, Week 66: number analyzed (Participants) | 38 | 4
  Chest Pain, Week 66 | -0.25 (0.92) | 0.25 (1.19)
  Chest Pain, Week 67: number analyzed (Participants) | 33 | 4
  Chest Pain, Week 67 | -0.18 (0.86) | 0.13 (1.44)
  Chest Pain, Week 68: number analyzed (Participants) | 34 | 4
  Chest Pain, Week 68 | -0.15 (0.93) | -0.25 (1.55)
  Chest Pain, Week 69: number analyzed (Participants) | 35 | 3
  Chest Pain, Week 69 | -0.13 (0.83) | -0.17 (1.89)
  Chest Pain, Week 70: number analyzed (Participants) | 36 | 3
  Chest Pain, Week 70 | -0.14 (0.93) | 0.00 (1.80)
  Chest Pain, Week 71: number analyzed (Participants) | 31 | 3
  Chest Pain, Week 71 | -0.10 (0.88) | 0.00 (0.87)
  Chest Pain, Week 72: number analyzed (Participants) | 29 | 2
  Chest Pain, Week 72 | -0.24 (0.85) | -1.00 (0.71)
  Chest Pain, Week 73: number analyzed (Participants) | 28 | 1
  Chest Pain, Week 73 | -0.25 (1.02) | -1.50
  Chest Pain, Week 74: number analyzed (Participants) | 31 | 1
  Chest Pain, Week 74 | -0.08 (0.93) | -1.50
  Chest Pain, Week 75: number analyzed (Participants) | 31 | 1
  Chest Pain, Week 75 | -0.21 (0.98) | -1.50
  Chest Pain, Week 76: number analyzed (Participants) | 29 | 1
  Chest Pain, Week 76 | 0.03 (1.00) | -1.50
  Chest Pain, Week 77: number analyzed (Participants) | 26 | 2
  Chest Pain, Week 77 | -0.06 (0.89) | -1.50 (0.00)
  Chest Pain, Week 78: number analyzed (Participants) | 23 | 1
  Chest Pain, Week 78 | -0.04 (0.84) | -1.50
  Chest Pain, Week 79: number analyzed (Participants) | 19 | 1
  Chest Pain, Week 79 | -0.11 (1.09) | -0.50
  Chest Pain, Week 80: number analyzed (Participants) | 20 | 1
  Chest Pain, Week 80 | -0.18 (1.05) | -1.50
  Chest Pain, Week 81: number analyzed (Participants) | 17 | 1
  Chest Pain, Week 81 | -0.59 (0.96) | -1.50
  Chest Pain, Week 82: number analyzed (Participants) | 18 | 1
  Chest Pain, Week 82 | -0.39 (0.96) | -1.50
  Chest Pain, Week 83: number analyzed (Participants) | 22 | 1
  Chest Pain, Week 83 | -0.34 (0.90) | -1.50
  Chest Pain, Week 84: number analyzed (Participants) | 20 | 1
  Chest Pain, Week 84 | -0.20 (0.75) | -1.50
  Chest Pain, Week 85: number analyzed (Participants) | 17 | 1
  Chest Pain, Week 85 | -0.44 (0.97) | -1.50
  Chest Pain, Week 86: number analyzed (Participants) | 12 | 1
  Chest Pain, Week 86 | -0.38 (0.64) | -1.50
  Chest Pain, Week 87: number analyzed (Participants) | 15 | 1
  Chest Pain, Week 87 | -0.53 (1.01) | -1.50
  Chest Pain, Week 88: number analyzed (Participants) | 14 | 1
  Chest Pain, Week 88 | -0.46 (1.06) | -1.50
  Chest Pain, Week 89: number analyzed (Participants) | 11 | 1
  Chest Pain, Week 89 | -0.55 (0.96) | -1.50
  Chest Pain, Week 90: number analyzed (Participants) | 14 | 1
  Chest Pain, Week 90 | -0.18 (0.85) | -1.50
  Chest Pain, Week 91: number analyzed (Participants) | 11 | 1
  Chest Pain, Week 91 | -0.32 (1.08) | -1.50
  Chest Pain, Week 92: number analyzed (Participants) | 10 | 1
  Chest Pain, Week 92 | -0.40 (0.66) | -1.50
  Chest Pain, Week 93: number analyzed (Participants) | 11 | 1
  Chest Pain, Week 93 | -0.18 (1.08) | -1.50
  Chest Pain, Week 94: number analyzed (Participants) | 10 | 0
  Chest Pain, Week 94 | -0.30 (1.09) |
  Chest Pain, Week 95: number analyzed (Participants) | 10 | 0
  Chest Pain, Week 95 | -0.05 (1.26) |
  Chest Pain, Week 96: number analyzed (Participants) | 9 | 0
  Chest Pain, Week 96 | -0.17 (1.25) |
  Chest Pain, Week 97: number analyzed (Participants) | 8 | 0
  Chest Pain, Week 97 | -0.19 (1.31) |
  Chest Pain, Week 98: number analyzed (Participants) | 10 | 0
  Chest Pain, Week 98 | -0.25 (1.16) |
  Chest Pain, Week 99: number analyzed (Participants) | 7 | 0
  Chest Pain, Week 99 | -0.21 (1.47) |
  Chest Pain, Week 100: number analyzed (Participants) | 6 | 0
  Chest Pain, Week 100 | -0.50 (1.38) |
  Chest Pain, Week 101: number analyzed (Participants) | 7 | 0
  Chest Pain, Week 101 | -0.36 (1.38) |
  Chest Pain, Week 102: number analyzed (Participants) | 4 | 0
  Chest Pain, Week 102 | -0.75 (1.71) |
  Chest Pain, Week 103: number analyzed (Participants) | 6 | 0
  Chest Pain, Week 103 | -0.33 (1.54) |
  Chest Pain, Week 104: number analyzed (Participants) | 5 | 0
  Chest Pain, Week 104 | -0.60 (1.39) |
  Chest Pain, Week 105: number analyzed (Participants) | 4 | 0
  Chest Pain, Week 105 | -1.00 (1.41) |
  Chest Pain, Week 106: number analyzed (Participants) | 4 | 0
  Chest Pain, Week 106 | -1.00 (1.41) |
  Chest Pain, Week 107: number analyzed (Participants) | 4 | 0
  Chest Pain, Week 107 | -1.00 (1.41) |
  Chest Pain, Week 108: number analyzed (Participants) | 4 | 0
  Chest Pain, Week 108 | -0.75 (1.50) |
  Chest Pain, Week 109: number analyzed (Participants) | 5 | 0
  Chest Pain, Week 109 | -0.60 (1.52) |
  Chest Pain, Week 110: number analyzed (Participants) | 6 | 0
  Chest Pain, Week 110 | -0.42 (1.43) |
  Chest Pain, Week 111: number analyzed (Participants) | 5 | 0
  Chest Pain, Week 111 | -0.50 (1.50) |
  Chest Pain, Week 112: number analyzed (Participants) | 4 | 0
  Chest Pain, Week 112 | -0.13 (0.63) |
  Chest Pain, Week 113: number analyzed (Participants) | 4 | 0
  Chest Pain, Week 113 | 0.13 (0.63) |
  Chest Pain, Week 114: number analyzed (Participants) | 3 | 0
  Chest Pain, Week 114 | 0.00 (1.00) |
  Chest Pain, Week 115: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 115 | 0.25 (0.35) |
  Chest Pain, Week 116: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 116 | 0.50 (0.71) |
  Chest Pain, Week 117: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 117 | 0.25 (1.06) |
  Chest Pain, Week 118: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 118 | -0.25 (1.06) |
  Chest Pain, Week 119: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 119 | -0.25 (0.35) |
  Chest Pain, Week 120: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 120 | 0.00 (0.71) |
  Chest Pain, Week 121: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 121 | 0.00 (1.41) |
  Chest Pain, Week 122: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 122 | 0.00 (1.41) |
  Chest Pain, Week 123: number analyzed (Participants) | 2 | 0
  Chest Pain, Week 123 | -0.75 (1.77) |
  Chest Pain, Week 124: number analyzed (Participants) | 1 | 0
  Chest Pain, Week 124 | 0.50 |
  Chest Pain, Week 125: number analyzed (Participants) | 1 | 0
  Chest Pain, Week 125 | 0.50 |
  Chest Pain, Survival Follow-Up Month 1: number analyzed (Participants) | 158 | 58
  Chest Pain, Survival Follow-Up Month 1 | 0.01 (1.13) | 0.22 (0.87)
  Chest Pain, Survival Follow-Up Month 2: number analyzed (Participants) | 42 | 47
  Chest Pain, Survival Follow-Up Month 2 | -0.07 (1.18) | -0.16 (0.96)
  Chest Pain, Survival Follow-Up Month 3: number analyzed (Participants) | 36 | 26
  Chest Pain, Survival Follow-Up Month 3 | 0.15 (1.33) | -0.08 (0.87)
  Chest Pain, Survival Follow-Up Month 4: number analyzed (Participants) | 23 | 28
  Chest Pain, Survival Follow-Up Month 4 | -0.28 (1.40) | -0.07 (0.79)
  Chest Pain, Survival Follow-Up Month 5: number analyzed (Participants) | 22 | 22
  Chest Pain, Survival Follow-Up Month 5 | -0.11 (1.49) | -0.02 (0.65)
  Chest Pain, Survival Follow-Up Month 6: number analyzed (Participants) | 15 | 21
  Chest Pain, Survival Follow-Up Month 6 | -0.37 (1.67) | 0.02 (0.78)
  Cough, Week 1: number analyzed (Participants) | 203 | 114
  Cough, Week 1 | 0.08 (0.69) | 0.04 (0.73)
  Cough, Week 2: number analyzed (Participants) | 204 | 108
  Cough, Week 2 | 0.02 (0.78) | 0.04 (0.84)
  Cough, Week 3: number analyzed (Participants) | 197 | 106
  Cough, Week 3 | 0.02 (0.86) | -0.09 (0.93)
  Cough, Week 4: number analyzed (Participants) | 190 | 102
  Cough, Week 4 | -0.06 (0.86) | -0.10 (0.93)
  Cough, Week 5: number analyzed (Participants) | 192 | 97
  Cough, Week 5 | -0.09 (0.84) | -0.09 (0.99)
  Cough, Week 6: number analyzed (Participants) | 182 | 98
  Cough, Week 6 | -0.15 (0.86) | -0.08 (0.98)
  Cough, Week 7: number analyzed (Participants) | 176 | 87
  Cough, Week 7 | -0.11 (0.86) | -0.06 (1.01)
  Cough, Week 8: number analyzed (Participants) | 169 | 80
  Cough, Week 8 | -0.13 (0.95) | -0.21 (1.04)
  Cough, Week 9: number analyzed (Participants) | 172 | 80
  Cough, Week 9 | -0.15 (0.99) | -0.13 (1.23)
  Cough, Week 10: number analyzed (Participants) | 166 | 75
  Cough, Week 10 | -0.20 (1.05) | -0.07 (1.17)
  Cough, Week 11: number analyzed (Participants) | 171 | 78
  Cough, Week 11 | -0.15 (1.03) | -0.15 (1.17)
  Cough, Week 12: number analyzed (Participants) | 160 | 72
  Cough, Week 12 | -0.17 (1.03) | -0.11 (1.09)
  Cough, Week 13: number analyzed (Participants) | 151 | 61
  Cough, Week 13 | -0.24 (1.08) | -0.04 (1.11)
  Cough, Week 14: number analyzed (Participants) | 144 | 62
  Cough, Week 14 | -0.23 (1.06) | -0.18 (1.08)
  Cough, Week 15: number analyzed (Participants) | 143 | 51
  Cough, Week 15 | -0.27 (1.06) | -0.05 (1.10)
  Cough, Week 16: number analyzed (Participants) | 139 | 52
  Cough, Week 16 | -0.37 (1.07) | -0.25 (1.09)
  Cough, Week 17: number analyzed (Participants) | 145 | 53
  Cough, Week 17 | -0.32 (1.09) | -0.21 (1.01)
  Cough, Week 18: number analyzed (Participants) | 136 | 49
  Cough, Week 18 | -0.33 (1.07) | -0.33 (1.09)
  Cough, Week 19: number analyzed (Participants) | 124 | 45
  Cough, Week 19 | -0.33 (1.06) | -0.40 (0.89)
  Cough, Week 20: number analyzed (Participants) | 123 | 43
  Cough, Week 20 | -0.37 (1.10) | -0.31 (0.90)
  Cough, Week 21: number analyzed (Participants) | 126 | 41
  Cough, Week 21 | -0.37 (1.08) | -0.33 (0.96)
  Cough, Week 22: number analyzed (Participants) | 116 | 37
  Cough, Week 22 | -0.37 (1.15) | -0.24 (0.97)
  Cough, Week 23: number analyzed (Participants) | 122 | 35
  Cough, Week 23 | -0.30 (1.10) | -0.41 (1.03)
  Cough, Week 24: number analyzed (Participants) | 110 | 34
  Cough, Week 24 | -0.38 (1.09) | -0.54 (1.04)
  Cough, Week 25: number analyzed (Participants) | 104 | 31
  Cough, Week 25 | -0.49 (0.91) | -0.47 (1.05)
  Cough, Week 26: number analyzed (Participants) | 109 | 31
  Cough, Week 26 | -0.43 (0.99) | -0.34 (1.02)
  Cough, Week 27: number analyzed (Participants) | 102 | 27
  Cough, Week 27 | -0.41 (0.97) | -0.48 (0.98)
  Cough, Week 28: number analyzed (Participants) | 96 | 28
  Cough, Week 28 | -0.52 (0.96) | -0.43 (0.84)
  Cough, Week 29: number analyzed (Participants) | 104 | 27
  Cough, Week 29 | -0.43 (0.98) | -0.46 (0.91)
  Cough, Week 30: number analyzed (Participants) | 100 | 23
  Cough, Week 30 | -0.43 (0.95) | -0.46 (1.07)
  Cough, Week 31: number analyzed (Participants) | 93 | 25
  Cough, Week 31 | -0.32 (1.07) | -0.38 (0.77)
  Cough, Week 32: number analyzed (Participants) | 88 | 25
  Cough, Week 32 | -0.30 (0.94) | -0.12 (0.99)
  Cough, Week 33: number analyzed (Participants) | 88 | 25
  Cough, Week 33 | -0.19 (1.12) | -0.52 (1.03)
  Cough, Week 34: number analyzed (Participants) | 85 | 24
  Cough, Week 34 | -0.35 (1.12) | -0.33 (1.03)
  Cough, Week 35: number analyzed (Participants) | 87 | 20
  Cough, Week 35 | -0.46 (1.01) | 0.00 (1.22)
  Cough, Week 36: number analyzed (Participants) | 85 | 20
  Cough, Week 36 | -0.35 (1.08) | -0.20 (1.01)
  Cough, Week 37: number analyzed (Participants) | 82 | 21
  Cough, Week 37 | -0.46 (1.03) | -0.45 (1.11)
  Cough, Week 38: number analyzed (Participants) | 83 | 19
  Cough, Week 38 | -0.38 (1.06) | -0.03 (0.89)
  Cough, Week 39: number analyzed (Participants) | 78 | 18
  Cough, Week 39 | -0.27 (0.99) | -0.17 (1.00)
  Cough, Week 40: number analyzed (Participants) | 76 | 14
  Cough, Week 40 | -0.38 (0.95) | -0.50 (0.90)
  Cough, Week 41: number analyzed (Participants) | 77 | 16
  Cough, Week 41 | -0.44 (0.92) | -0.22 (0.77)
  Cough, Week 42: number analyzed (Participants) | 70 | 16
  Cough, Week 42 | -0.44 (0.92) | -0.41 (0.97)
  Cough, Week 43: number analyzed (Participants) | 68 | 16
  Cough, Week 43 | -0.39 (0.98) | -0.13 (0.92)
  Cough, Week 44: number analyzed (Participants) | 76 | 16
  Cough, Week 44 | -0.38 (0.94) | -0.16 (0.89)
  Cough, Week 45: number analyzed (Participants) | 69 | 14
  Cough, Week 45 | -0.30 (1.10) | -0.14 (1.03)
  Cough, Week 46: number analyzed (Participants) | 71 | 15
  Cough, Week 46 | -0.25 (0.99) | -0.03 (1.23)
  Cough, Week 47: number analyzed (Participants) | 70 | 13
  Cough, Week 47 | -0.44 (0.88) | -0.12 (1.23)
  Cough, Week 48: number analyzed (Participants) | 66 | 11
  Cough, Week 48 | -0.29 (0.99) | 0.14 (1.21)
  Cough, Week 49: number analyzed (Participants) | 65 | 9
  Cough, Week 49 | -0.38 (1.00) | -0.56 (1.36)
  Cough, Week 50: number analyzed (Participants) | 70 | 8
  Cough, Week 50 | -0.39 (0.96) | -0.19 (1.16)
  Cough, Week 51: number analyzed (Participants) | 65 | 10
  Cough, Week 51 | -0.30 (1.00) | -0.40 (1.20)
  Cough, Week 52: number analyzed (Participants) | 72 | 7
  Cough, Week 52 | -0.32 (1.03) | -0.21 (1.07)
  Cough, Week 53: number analyzed (Participants) | 64 | 6
  Cough, Week 53 | -0.37 (1.03) | -0.17 (1.33)
  Cough, Week 54: number analyzed (Participants) | 65 | 7
  Cough, Week 54 | -0.41 (0.93) | -0.07 (1.21)
  Cough, Week 55: number analyzed (Participants) | 62 | 5
  Cough, Week 55 | -0.40 (0.93) | 0.10 (1.34)
  Cough, Week 56: number analyzed (Participants) | 62 | 6
  Cough, Week 56 | -0.26 (0.94) | 0.17 (1.13)
  Cough, Week 57: number analyzed (Participants) | 62 | 5
  Cough, Week 57 | -0.35 (0.98) | 0.00 (1.27)
  Cough, Week 58: number analyzed (Participants) | 56 | 4
  Cough, Week 58 | -0.33 (1.06) | 0.13 (1.31)
  Cough, Week 59: number analyzed (Participants) | 52 | 4
  Cough, Week 59 | -0.31 (0.97) | 0.13 (1.60)
  Cough, Week 60: number analyzed (Participants) | 48 | 4
  Cough, Week 60 | -0.42 (0.89) | 0.38 (1.18)
  Cough, Week 61: number analyzed (Participants) | 49 | 5
  Cough, Week 61 | -0.35 (0.95) | 0.80 (1.20)
  Cough, Week 62: number analyzed (Participants) | 41 | 5
  Cough, Week 62 | -0.23 (1.03) | 0.50 (1.62)
  Cough, Week 63: number analyzed (Participants) | 43 | 5
  Cough, Week 63 | -0.22 (1.04) | 0.50 (1.27)
  Cough, Week 64: number analyzed (Participants) | 42 | 4
  Cough, Week 64 | -0.19 (1.07) | 0.00 (1.87)
  Cough, Week 65: number analyzed (Participants) | 40 | 3
  Cough, Week 65 | -0.23 (1.04) | 0.83 (1.04)
  Cough, Week 66: number analyzed (Participants) | 38 | 4
  Cough, Week 66 | -0.29 (0.90) | 0.63 (1.03)
  Cough, Week 67: number analyzed (Participants) | 33 | 4
  Cough, Week 67 | -0.48 (0.91) | 0.38 (1.38)
  Cough, Week 68: number analyzed (Participants) | 34 | 4
  Cough, Week 68 | -0.34 (0.82) | 0.13 (1.49)
  Cough, Week 69: number analyzed (Participants) | 35 | 3
  Cough, Week 69 | -0.34 (1.03) | 0.17 (1.61)
  Cough, Week 70: number analyzed (Participants) | 36 | 3
  Cough, Week 70 | -0.26 (0.94) | 0.17 (1.61)
  Cough, Week 71: number analyzed (Participants) | 31 | 3
  Cough, Week 71 | -0.23 (0.91) | 0.33 (1.04)
  Cough, Week 72: number analyzed (Participants) | 29 | 2
  Cough, Week 72 | -0.48 (0.87) | -1.50 (1.41)
  Cough, Week 73: number analyzed (Participants) | 28 | 1
  Cough, Week 73 | -0.43 (0.91) | -0.50
  Cough, Week 74: number analyzed (Participants) | 31 | 1
  Cough, Week 74 | -0.42 (0.93) | -0.50
  Cough, Week 75: number analyzed (Participants) | 31 | 1
  Cough, Week 75 | -0.32 (1.00) | -0.50
  Cough, Week 76: number analyzed (Participants) | 29 | 1
  Cough, Week 76 | -0.31 (0.91) | -0.50
  Cough, Week 77: number analyzed (Participants) | 26 | 2
  Cough, Week 77 | -0.40 (0.92) | -0.50 (2.83)
  Cough, Week 78: number analyzed (Participants) | 23 | 1
  Cough, Week 78 | -0.52 (0.94) | 0.00
  Cough, Week 79: number analyzed (Participants) | 19 | 1
  Cough, Week 79 | -0.08 (0.93) | 1.00
  Cough, Week 80: number analyzed (Participants) | 20 | 1
  Cough, Week 80 | -0.48 (0.87) | 1.00
  Cough, Week 81: number analyzed (Participants) | 17 | 1
  Cough, Week 81 | -0.44 (1.01) | -0.50
  Cough, Week 82: number analyzed (Participants) | 18 | 1
  Cough, Week 82 | -0.39 (0.90) | 1.00
  Cough, Week 83: number analyzed (Participants) | 22 | 1
  Cough, Week 83 | -0.25 (1.09) | 0.50
  Cough, Week 84: number analyzed (Participants) | 20 | 1
  Cough, Week 84 | -0.30 (0.91) | 1.00
  Cough, Week 85: number analyzed (Participants) | 17 | 1
  Cough, Week 85 | -0.32 (1.25) | 1.50
  Cough, Week 86: number analyzed (Participants) | 12 | 1
  Cough, Week 86 | -0.54 (1.27) | 0.00
  Cough, Week 87: number analyzed (Participants) | 15 | 1
  Cough, Week 87 | -0.33 (1.18) | 0.00
  Cough, Week 88: number analyzed (Participants) | 14 | 1
  Cough, Week 88 | -0.46 (1.26) | 0.00
  Cough, Week 89: number analyzed (Participants) | 11 | 1
  Cough, Week 89 | -0.36 (1.07) | 0.00
  Cough, Week 90: number analyzed (Participants) | 14 | 1
  Cough, Week 90 | -0.29 (1.05) | 0.00
  Cough, Week 91: number analyzed (Participants) | 11 | 1
  Cough, Week 91 | -0.27 (1.17) | 0.00
  Cough, Week 92: number analyzed (Participants) | 10 | 1
  Cough, Week 92 | -0.35 (1.27) | 1.00
  Cough, Week 93: number analyzed (Participants) | 11 | 1
  Cough, Week 93 | -0.55 (0.96) | 0.00
  Cough, Week 94: number analyzed (Participants) | 10 | 0
  Cough, Week 94 | -0.40 (0.81) |
  Cough, Week 95: number analyzed (Participants) | 10 | 0
  Cough, Week 95 | 0.05 (1.23) |
  Cough, Week 96: number analyzed (Participants) | 9 | 0
  Cough, Week 96 | -0.28 (1.28) |
  Cough, Week 97: number analyzed (Participants) | 8 | 0
  Cough, Week 97 | -0.31 (1.19) |
  Cough, Week 98: number analyzed (Participants) | 10 | 0
  Cough, Week 98 | -0.10 (0.99) |
  Cough, Week 99: number analyzed (Participants) | 7 | 0
  Cough, Week 99 | -0.43 (0.98) |
  Cough, Week 100: number analyzed (Participants) | 6 | 0
  Cough, Week 100 | -0.58 (0.86) |
  Cough, Week 101: number analyzed (Participants) | 7 | 0
  Cough, Week 101 | -0.50 (0.96) |
  Cough, Week 102: number analyzed (Participants) | 4 | 0
  Cough, Week 102 | -0.50 (0.41) |
  Cough, Week 103: number analyzed (Participants) | 6 | 0
  Cough, Week 103 | -0.75 (0.42) |
  Cough, Week 104: number analyzed (Participants) | 5 | 0
  Cough, Week 104 | -0.80 (0.27) |
  Cough, Week 105: number analyzed (Participants) | 4 | 0
  Cough, Week 105 | -0.63 (0.48) |
  Cough, Week 106: number analyzed (Participants) | 4 | 0
  Cough, Week 106 | -0.63 (0.48) |
  Cough, Week 107: number analyzed (Participants) | 4 | 0
  Cough, Week 107 | -0.63 (0.48) |
  Cough, Week 108: number analyzed (Participants) | 4 | 0
  Cough, Week 108 | -0.50 (0.71) |
  Cough, Week 109: number analyzed (Participants) | 5 | 0
  Cough, Week 109 | -0.50 (0.50) |
  Cough, Week 110: number analyzed (Participants) | 6 | 0
  Cough, Week 110 | -0.50 (0.45) |
  Cough, Week 111: number analyzed (Participants) | 5 | 0
  Cough, Week 111 | -0.30 (0.84) |
  Cough, Week 112: number analyzed (Participants) | 4 | 0
  Cough, Week 112 | -0.63 (0.48) |
  Cough, Week 113: number analyzed (Participants) | 4 | 0
  Cough, Week 113 | -0.25 (0.65) |
  Cough, Week 114: number analyzed (Participants) | 3 | 0
  Cough, Week 114 | -0.33 (0.29) |
  Cough, Week 115: number analyzed (Participants) | 2 | 0
  Cough, Week 115 | 0.25 (0.35) |
  Cough, Week 116: number analyzed (Participants) | 2 | 0
  Cough, Week 116 | -0.25 (1.06) |
  Cough, Week 117: number analyzed (Participants) | 2 | 0
  Cough, Week 117 | -0.50 (0.71) |
  Cough, Week 118: number analyzed (Participants) | 2 | 0
  Cough, Week 118 | -0.25 (0.35) |
  Cough, Week 119: number analyzed (Participants) | 2 | 0
  Cough, Week 119 | 0.00 (0.00) |
  Cough, Week 120: number analyzed (Participants) | 2 | 0
  Cough, Week 120 | -0.25 (0.35) |
  Cough, Week 121: number analyzed (Participants) | 2 | 0
  Cough, Week 121 | -0.50 (0.71) |
  Cough, Week 122: number analyzed (Participants) | 2 | 0
  Cough, Week 122 | -0.50 (0.71) |
  Cough, Week 123: number analyzed (Participants) | 2 | 0
  Cough, Week 123 | -0.75 (1.06) |
  Cough, Week 124: number analyzed (Participants) | 1 | 0
  Cough, Week 124 | 0.50 |
  Cough, Week 125: number analyzed (Participants) | 1 | 0
  Cough, Week 125 | 0.50 |
  Cough, Survival Follow-Up Month 1: number analyzed (Participants) | 158 | 58
  Cough, Survival Follow-Up Month 1 | -0.21 (1.05) | -0.01 (0.96)
  Cough, Survival Follow-Up Month 2: number analyzed (Participants) | 42 | 47
  Cough, Survival Follow-Up Month 2 | -0.07 (1.16) | -0.31 (1.18)
  Cough, Survival Follow-Up Month 3: number analyzed (Participants) | 36 | 26
  Cough, Survival Follow-Up Month 3 | -0.14 (1.12) | -0.13 (1.32)
  Cough, Survival Follow-Up Month 4: number analyzed (Participants) | 23 | 28
  Cough, Survival Follow-Up Month 4 | -0.39 (1.15) | -0.45 (1.17)
  Cough, Survival Follow-Up Month 5: number analyzed (Participants) | 22 | 22
  Cough, Survival Follow-Up Month 5 | -0.25 (1.44) | -0.27 (1.32)
  Cough, Survival Follow-Up Month 6: number analyzed (Participants) | 15 | 21
  Cough, Survival Follow-Up Month 6 | -0.23 (1.53) | -0.29 (1.26)
  Dyspnoea, Week 1: number analyzed (Participants) | 203 | 114
  Dyspnoea, Week 1 | 0.13 (0.76) | 0.23 (0.79)
  Dyspnoea, Week 2: number analyzed (Participants) | 204 | 108
  Dyspnoea, Week 2 | 0.10 (0.68) | 0.31 (0.84)
  Dyspnoea, Week 3: number analyzed (Participants) | 197 | 106
  Dyspnoea, Week 3 | 0.22 (0.78) | 0.32 (0.76)
  Dyspnoea, Week 4: number analyzed (Participants) | 190 | 102
  Dyspnoea, Week 4 | 0.23 (0.80) | 0.45 (0.84)
  Dyspnoea, Week 5: number analyzed (Participants) | 192 | 97
  Dyspnoea, Week 5 | 0.26 (0.84) | 0.42 (0.92)
  Dyspnoea, Week 6: number analyzed (Participants) | 182 | 96
  Dyspnoea, Week 6 | 0.27 (0.92) | 0.51 (0.95)
  Dyspnoea, Week 7: number analyzed (Participants) | 176 | 87
  Dyspnoea, Week 7 | 0.29 (0.88) | 0.60 (1.00)
  Dyspnoea, Week 8: number analyzed (Participants) | 169 | 80
  Dyspnoea, Week 8 | 0.32 (0.97) | 0.53 (1.02)
  Dyspnoea, Week 9: number analyzed (Participants) | 172 | 80
  Dyspnoea, Week 9 | 0.38 (0.95) | 0.62 (1.07)
  Dyspnoea, Week 10: number analyzed (Participants) | 166 | 75
  Dyspnoea, Week 10 | 0.41 (1.04) | 0.75 (1.13)
  Dyspnoea, Week 11: number analyzed (Participants) | 171 | 78
  Dyspnoea, Week 11 | 0.50 (1.05) | 0.60 (1.06)
  Dyspnoea, Week 12: number analyzed (Participants) | 160 | 72
  Dyspnoea, Week 12 | 0.47 (1.07) | 0.74 (1.08)
  Dyspnoea, Week 13: number analyzed (Participants) | 151 | 61
  Dyspnoea, Week 13 | 0.32 (1.00) | 0.76 (1.00)
  Dyspnoea, Week 14: number analyzed (Participants) | 144 | 62
  Dyspnoea, Week 14 | 0.34 (0.99) | 0.61 (1.10)
  Dyspnoea, Week 15: number analyzed (Participants) | 143 | 51
  Dyspnoea, Week 15 | 0.29 (1.06) | 0.71 (1.02)
  Dyspnoea, Week 16: number analyzed (Participants) | 139 | 52
  Dyspnoea, Week 16 | 0.22 (0.99) | 0.67 (1.11)
  Dyspnoea, Week 17: number analyzed (Participants) | 145 | 53
  Dyspnoea, Week 17 | 0.28 (1.10) | 0.68 (1.03)
  Dyspnoea, Week 18: number analyzed (Participants) | 136 | 49
  Dyspnoea, Week 18 | 0.23 (1.02) | 0.62 (1.03)
  Dyspnoea, Week 19: number analyzed (Participants) | 124 | 45
  Dyspnoea, Week 19 | 0.26 (1.06) | 0.54 (0.95)
  Dyspnoea, Week 20: number analyzed (Participants) | 123 | 43
  Dyspnoea, Week 20 | 0.24 (1.02) | 0.54 (1.08)
  Dyspnoea, Week 21: number analyzed (Participants) | 126 | 41
  Dyspnoea, Week 21 | 0.26 (1.04) | 0.39 (1.05)
  Dyspnoea, Week 22: number analyzed (Participants) | 116 | 37
  Dyspnoea, Week 22 | 0.21 (0.94) | 0.41 (1.05)
  Dyspnoea, Week 23: number analyzed (Participants) | 122 | 35
  Dyspnoea, Week 23 | 0.18 (0.97) | 0.41 (1.06)
  Dyspnoea, Week 24: number analyzed (Participants) | 110 | 34
  Dyspnoea, Week 24 | 0.22 (0.93) | 0.31 (1.01)
  Dyspnoea, Week 25: number analyzed (Participants) | 104 | 31
  Dyspnoea, Week 25 | 0.21 (0.88) | 0.20 (0.91)
  Dyspnoea, Week 26: number analyzed (Participants) | 109 | 31
  Dyspnoea, Week 26 | 0.17 (0.89) | 0.30 (1.00)
  Dyspnoea, Week 27: number analyzed (Participants) | 102 | 27
  Dyspnoea, Week 27 | 0.20 (1.04) | 0.30 (0.92)
  Dyspnoea, Week 28: number analyzed (Participants) | 96 | 28
  Dyspnoea, Week 28 | 0.16 (0.94) | 0.22 (1.01)
  Dyspnoea, Week 29: number analyzed (Participants) | 104 | 27
  Dyspnoea, Week 29 | 0.16 (0.92) | 0.33 (0.98)
  Dyspnoea, Week 30: number analyzed (Participants) | 100 | 23
  Dyspnoea, Week 30 | 0.24 (1.04) | 0.27 (1.02)
  Dyspnoea, Week 31: number analyzed (Participants) | 93 | 25
  Dyspnoea, Week 31 | 0.12 (0.99) | 0.26 (1.04)
  Dyspnoea, Week 32: number analyzed (Participants) | 88 | 25
  Dyspnoea, Week 32 | 0.20 (0.95) | 0.38 (1.06)
  Dyspnoea, Week 33: number analyzed (Participants) | 88 | 25
  Dyspnoea, Week 33 | 0.18 (0.98) | 0.19 (1.14)
  Dyspnoea, Week 34: number analyzed (Participants) | 85 | 24
  Dyspnoea, Week 34 | 0.21 (1.06) | 0.30 (1.02)
  Dyspnoea, Week 35: number analyzed (Participants) | 87 | 20
  Dyspnoea, Week 35 | 0.22 (1.03) | 0.46 (0.96)
  Dyspnoea, Week 36: number analyzed (Participants) | 85 | 20
  Dyspnoea, Week 36 | 0.21 (1.09) | 0.34 (1.14)
  Dyspnoea, Week 37: number analyzed (Participants) | 82 | 21
  Dyspnoea, Week 37 | 0.16 (1.13) | 0.10 (1.07)
  Dyspnoea, Week 38: number analyzed (Participants) | 83 | 19
  Dyspnoea, Week 38 | 0.18 (1.07) | 0.51 (0.99)
  Dyspnoea, Week 39: number analyzed (Participants) | 78 | 18
  Dyspnoea, Week 39 | 0.31 (1.04) | 0.26 (0.83)
  Dyspnoea, Week 40: number analyzed (Participants) | 76 | 14
  Dyspnoea, Week 40 | 0.31 (0.99) | 0.04 (0.79)
  Dyspnoea, Week 41: number analyzed (Participants) | 77 | 16
  Dyspnoea, Week 41 | 0.24 (0.99) | 0.18 (0.85)
  Dyspnoea, Week 42: number analyzed (Participants) | 70 | 16
  Dyspnoea, Week 42 | 0.26 (1.03) | 0.08 (0.70)
  Dyspnoea, Week 43: number analyzed (Participants) | 68 | 16
  Dyspnoea, Week 43 | 0.17 (1.13) | 0.41 (0.91)
  Dyspnoea, Week 44: number analyzed (Participants) | 76 | 16
  Dyspnoea, Week 44 | 0.22 (1.06) | 0.29 (0.86)
  Dyspnoea, Week 45: number analyzed (Participants) | 69 | 14
  Dyspnoea, Week 45 | 0.26 (1.09) | 0.31 (0.90)
  Dyspnoea, Week 46: number analyzed (Participants) | 71 | 15
  Dyspnoea, Week 46 | 0.29 (0.99) | 0.47 (1.03)
  Dyspnoea, Week 47: number analyzed (Participants) | 70 | 13
  Dyspnoea, Week 47 | 0.20 (1.02) | 0.45 (0.85)
  Dyspnoea, Week 48: number analyzed (Participants) | 66 | 11
  Dyspnoea, Week 48 | 0.32 (1.00) | 0.29 (0.91)
  Dyspnoea, Week 49: number analyzed (Participants) | 65 | 9
  Dyspnoea, Week 49 | 0.24 (1.04) | 0.00 (1.30)
  Dyspnoea, Week 50: number analyzed (Participants) | 70 | 8
  Dyspnoea, Week 50 | 0.32 (0.98) | 0.43 (0.88)
  Dyspnoea, Week 51: number analyzed (Participants) | 65 | 10
  Dyspnoea, Week 51 | 0.24 (0.92) | 0.06 (1.04)
  Dyspnoea, Week 52: number analyzed (Participants) | 72 | 7
  Dyspnoea, Week 52 | 0.27 (0.95) | 0.29 (0.90)
  Dyspnoea, Week 53: number analyzed (Participants) | 64 | 6
  Dyspnoea, Week 53 | 0.24 (1.00) | 0.30 (0.85)
  Dyspnoea, Week 54: number analyzed (Participants) | 65 | 7
  Dyspnoea, Week 54 | 0.28 (0.89) | 0.40 (0.95)
  Dyspnoea, Week 55: number analyzed (Participants) | 62 | 5
  Dyspnoea, Week 55 | 0.26 (0.98) | 0.44 (1.02)
  Dyspnoea, Week 56: number analyzed (Participants) | 62 | 6
  Dyspnoea, Week 56 | 0.26 (0.97) | 0.53 (1.10)
  Dyspnoea, Week 57: number analyzed (Participants) | 62 | 5
  Dyspnoea, Week 57 | 0.37 (0.95) | 0.24 (1.08)
  Dyspnoea, Week 58: number analyzed (Participants) | 56 | 4
  Dyspnoea, Week 58 | 0.19 (1.01) | 0.35 (1.40)
  Dyspnoea, Week 59: number analyzed (Participants) | 52 | 4
  Dyspnoea, Week 59 | 0.32 (0.84) | 0.35 (1.40)
  Dyspnoea, Week 60: number analyzed (Participants) | 48 | 4
  Dyspnoea, Week 60 | 0.35 (0.99) | 0.50 (1.51)
  Dyspnoea, Week 61: number analyzed (Participants) | 49 | 5
  Dyspnoea, Week 61 | 0.33 (1.03) | 0.60 (1.40)
  Dyspnoea, Week 62: number analyzed (Participants) | 41 | 5
  Dyspnoea, Week 62 | 0.45 (0.99) | 0.72 (1.36)
  Dyspnoea, Week 63: number analyzed (Participants) | 43 | 5
  Dyspnoea, Week 63 | 0.44 (1.05) | 0.56 (1.35)
  Dyspnoea, Week 64: number analyzed (Participants) | 42 | 4
  Dyspnoea, Week 64 | 0.36 (0.98) | -0.50 (1.91)
  Dyspnoea, Week 65: number analyzed (Participants) | 40 | 3
  Dyspnoea, Week 65 | 0.27 (0.97) | 0.07 (1.68)
  Dyspnoea, Week 66: number analyzed (Participants) | 38 | 4
  Dyspnoea, Week 66 | 0.32 (1.11) | 0.50 (1.23)
  Dyspnoea, Week 67: number analyzed (Participants) | 33 | 4
  Dyspnoea, Week 67 | 0.28 (0.91) | 0.40 (1.36)
  Dyspnoea, Week 68: number analyzed (Participants) | 34 | 4
  Dyspnoea, Week 68 | 0.35 (0.96) | 0.40 (1.43)
  Dyspnoea, Week 69: number analyzed (Participants) | 35 | 3
  Dyspnoea, Week 69 | 0.44 (1.02) | 0.73 (1.55)
  Dyspnoea, Week 70: number analyzed (Participants) | 36 | 3
  Dyspnoea, Week 70 | 0.33 (0.97) | 0.73 (1.55)
  Dyspnoea, Week 71: number analyzed (Participants) | 31 | 3
  Dyspnoea, Week 71 | 0.50 (0.95) | 0.60 (1.51)
  Dyspnoea, Week 72: number analyzed (Participants) | 29 | 3
  Dyspnoea, Week 72 | 0.17 (0.95) | 0.60 (1.44)
  Dyspnoea, Week 73: number analyzed (Participants) | 28 | 2
  Dyspnoea, Week 73 | 0.41 (0.96) | -1.80 (1.13)
  Dyspnoea, Week 74: number analyzed (Participants) | 31 | 1
  Dyspnoea, Week 74 | 0.30 (1.00) | -1.00
  Dyspnoea, Week 75: number analyzed (Participants) | 31 | 1
  Dyspnoea, Week 75 | 0.26 (0.89) | -1.00
  Dyspnoea, Week 76: number analyzed (Participants) | 29 | 1
  Dyspnoea, Week 76 | 0.23 (0.89) | -1.00
  Dyspnoea, Week 77: number analyzed (Participants) | 26 | 2
  Dyspnoea, Week 77 | 0.20 (0.97) | -1.50 (1.56)
  Dyspnoea, Week 78: number analyzed (Participants) | 23 | 1
  Dyspnoea, Week 78 | 0.31 (0.94) | -1.00
  Dyspnoea, Week 79: number analyzed (Participants) | 19 | 1
  Dyspnoea, Week 79 | 0.32 (0.95) | -1.00
  Dyspnoea, Week 80: number analyzed (Participants) | 20 | 1
  Dyspnoea, Week 80 | 0.30 (0.92) | -1.00
  Dyspnoea, Week 81: number analyzed (Participants) | 17 | 1
  Dyspnoea, Week 81 | -0.12 (1.00) | -0.80
  Dyspnoea, Week 82: number analyzed (Participants) | 18 | 1
  Dyspnoea, Week 82 | 0.02 (1.06) | -0.80
  Dyspnoea, Week 83: number analyzed (Participants) | 22 | 1
  Dyspnoea, Week 83 | 0.13 (1.01) | -1.00
  Dyspnoea, Week 84: number analyzed (Participants) | 20 | 1
  Dyspnoea, Week 84 | 0.19 (1.00) | -1.00
  Dyspnoea, Week 85: number analyzed (Participants) | 17 | 1
  Dyspnoea, Week 85 | 0.05 (1.17) | -0.80
  Dyspnoea, Week 86: number analyzed (Participants) | 12 | 1
  Dyspnoea, Week 86 | -0.07 (1.05) | -1.00
  Dyspnoea, Week 87: number analyzed (Participants) | 15 | 1
  Dyspnoea, Week 87 | -0.11 (0.96) | -1.00
  Dyspnoea, Week 88: number analyzed (Participants) | 14 | 1
  Dyspnoea, Week 88 | 0.06 (1.12) | -1.00
  Dyspnoea, Week 89: number analyzed (Participants) | 11 | 1
  Dyspnoea, Week 89 | 0.09 (0.91) | -1.00
  Dyspnoea, Week 90: number analyzed (Participants) | 14 | 1
  Dyspnoea, Week 90 | 0.37 (0.83) | -1.00
  Dyspnoea, Week 91: number analyzed (Participants) | 11 | 1
  Dyspnoea, Week 91 | 0.33 (1.11) | -1.00
  Dyspnoea, Week 92: number analyzed (Participants) | 10 | 1
  Dyspnoea, Week 92 | 0.20 (1.05) | -0.80
  Dyspnoea, Week 93: number analyzed (Participants) | 11 | 1
  Dyspnoea, Week 93 | 0.35 (0.96) | -0.80
  Dyspnoea, Week 94: number analyzed (Participants) | 10 | 0
  Dyspnoea, Week 94 | 0.50 (0.93) |
  Dyspnoea, Week 95: number analyzed (Participants) | 10 | 0
  Dyspnoea, Week 95 | 0.48 (0.98) |
  Dyspnoea, Week 96: number analyzed (Participants) | 9 | 0
  Dyspnoea, Week 96 | 0.51 (1.09) |
  Dyspnoea, Week 97: number analyzed (Participants) | 8 | 0
  Dyspnoea, Week 97 | 0.33 (1.18) |
  Dyspnoea, Week 98: number analyzed (Participants) | 10 | 0
  Dyspnoea, Week 98 | 0.38 (1.05) |
  Dyspnoea, Week 99: number analyzed (Participants) | 7 | 0
  Dyspnoea, Week 99 | 0.11 (0.99) |
  Dyspnoea, Week 100: number analyzed (Participants) | 6 | 0
  Dyspnoea, Week 100 | 0.27 (1.11) |
  Dyspnoea, Week 101: number analyzed (Participants) | 7 | 0
  Dyspnoea, Week 101 | 0.20 (1.11) |
  Dyspnoea, Week 102: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 102 | 0.35 (1.06) |
  Dyspnoea, Week 103: number analyzed (Participants) | 6 | 0
  Dyspnoea, Week 103 | 0.47 (1.29) |
  Dyspnoea, Week 104: number analyzed (Participants) | 5 | 0
  Dyspnoea, Week 104 | 0.48 (1.22) |
  Dyspnoea, Week 105: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 105 | -0.20 (0.71) |
  Dyspnoea, Week 106: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 106 | -0.20 (0.99) |
  Dyspnoea, Week 107: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 107 | -0.30 (0.62) |
  Dyspnoea, Week 108: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 108 | -0.15 (0.98) |
  Dyspnoea, Week 109: number analyzed (Participants) | 5 | 0
  Dyspnoea, Week 109 | 0.16 (1.17) |
  Dyspnoea, Week 110: number analyzed (Participants) | 6 | 0
  Dyspnoea, Week 110 | 0.33 (1.00) |
  Dyspnoea, Week 111: number analyzed (Participants) | 5 | 0
  Dyspnoea, Week 111 | -0.04 (0.86) |
  Dyspnoea, Week 112: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 112 | 0.20 (0.43) |
  Dyspnoea, Week 113: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 113 | 0.20 (0.67) |
  Dyspnoea, Week 114: number analyzed (Participants) | 3 | 0
  Dyspnoea, Week 114 | 0.40 (0.72) |
  Dyspnoea, Week 115: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 115 | 0.80 (0.85) |
  Dyspnoea, Week 116: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 116 | 0.60 (0.57) |
  Dyspnoea, Week 117: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 117 | 0.30 (0.14) |
  Dyspnoea, Week 118: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 118 | 0.30 (0.42) |
  Dyspnoea, Week 119: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 119 | 0.50 (0.42) |
  Dyspnoea, Week 120: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 120 | 0.30 (0.42) |
  Dyspnoea, Week 121: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 121 | 0.60 (0.57) |
  Dyspnoea, Week 122: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 122 | 0.60 (0.00) |
  Dyspnoea, Week 123: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 123 | -0.20 (0.57) |
  Dyspnoea, Week 124: number analyzed (Participants) | 1 | 0
  Dyspnoea, Week 124 | -0.20 |
  Dyspnoea, Week 125: number analyzed (Participants) | 1 | 0
  Dyspnoea, Week 125 | 0.20 |
  Dyspnoea, Survival Follow-Up Month 1: number analyzed (Participants) | 158 | 58
  Dyspnoea, Survival Follow-Up Month 1 | 0.41 (1.11) | 0.60 (1.14)
  Dyspnoea, Survival Follow-Up Month 2: number analyzed (Participants) | 42 | 47
  Dyspnoea, Survival Follow-Up Month 2 | 0.36 (1.20) | 0.46 (1.22)
  Dyspnoea, Survival Follow-Up Month 3: number analyzed (Participants) | 36 | 26
  Dyspnoea, Survival Follow-Up Month 3 | 0.27 (0.96) | 0.61 (1.19)
  Dyspnoea, Survival Follow-Up Month 4: number analyzed (Participants) | 23 | 28
  Dyspnoea, Survival Follow-Up Month 4 | 0.02 (1.11) | 0.45 (0.88)
  Dyspnoea, Survival Follow-Up Month 5: number analyzed (Participants) | 22 | 22
  Dyspnoea, Survival Follow-Up Month 5 | 0.13 (1.24) | 0.48 (1.00)
  Dyspnoea, Survival Follow-Up Month 6: number analyzed (Participants) | 15 | 21
  Dyspnoea, Survival Follow-Up Month 6 | -0.09 (1.29) | 0.54 (0.97)

13. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with at least one adverse event. Adverse event onset date before cross over.
Time Frame: Up to approximately 69 months after first patient enrolled
Population: The safety-evaluable population included all treated participants, defined as randomized participants who received any protocol treatment. For the safety analyses, participants were grouped according to whether any full or partial dose of atezolizumab was received, including when atezolizumab was received in error. Specifically, for participants randomized to the CnP arm, if atezolizumab was received in error, the participants were grouped to the Atezo+CnP arm for the safety analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 473 | 232
Percentage of participants | 99.6 | 98.7

14. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezolizumab
Description: Baseline prevalence and post-baseline incidence of anti-drug antibodies (ADA) to Atezolizumab in the Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed) and Arm B Carboplatin+nab-paclitaxel Crossover Participants
Time Frame: Up to approximately 35 months after first subject enrolled
Population: The baseline ADA-evaluable population included participants who had a baseline ADA result. The post-baseline ADA-evaluable population included participants who had at least one post-baseline ADA result and who had received at least one dose of study treatment. The ADA-evaluable WT population was defined as the ADA-evaluable population excluding participants with an activating EGFR mutation or ALK translocation.
Measure: Number; unit: Perecentage of participants
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 473 | 96
Perecentage of participants
  Baseline: number analyzed (Participants) | 473 | 84
  Baseline | 3.1 | 4.8
  Post-baseline: number analyzed (Participants) | 446 | 96
  Post-baseline | 22.4 | 23.5

15. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Atezolizumab for Patients in Atezolizumab+Carboplatin+Nab-Paclitaxel Arm
Description: Predose samples will be collected on the same day of treatment administration. The infusion duration of atezolizumab will be of 30-60 minutes.
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1 (Cycle length = 21 days)
Population: The PK-evaluable population was defined as all participants who received any dose of atezolizumab, carboplatin, or nab-paclitaxel and who had evaluable PK samples.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 465
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 437
  Cycle 1 Day 1 | 392 (114)
  Cycle 3 Day 1: number analyzed (Participants) | 356
  Cycle 3 Day 1 | 454 (170)

16. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Atezolizumab Prior to Infusion in Atezolizumab+Carboplain+Nab-Paclitaxel
Description: Predose samples will be collected on the same day of treatment administration.
Time Frame: Cycle 1 Day 21, Cycle 2 Day 21, Cycle 3 Day 21, and Cycle 7 Day 21 (Cycle length = 21 days)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin)
Number analyzed (Participants) | 465
mcg/mL
  Cycle 1 Day 21: number analyzed (Participants) | 416
  Cycle 1 Day 21 | 70.9 (35.1)
  Cycle 2 Day 21: number analyzed (Participants) | 384
  Cycle 2 Day 21 | 111 (52.2)
  Cycle 3 Day 21: number analyzed (Participants) | 352
  Cycle 3 Day 21 | 134 (57.8)
  Cycle 7 Day 21: number analyzed (Participants) | 257
  Cycle 7 Day 21 | 218 (93.7)

17. Secondary Outcome: Plasma Concentrations of Carboplatin
Time Frame: Predose (same day of treatment administration), 5-10 minutes before end of carboplatin infusion, 1 hour after carboplatin infusion (infusion duration=15 to 30 minutes) on Day 1 of Cycle 1 and 3 (1 Cycle=21 days) (up to approximately 35 months)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Arm B (Nab-Paclitaxel+Carboplatin Crossover): Participants received IV infusion of carboplatin on Day 1 and nab-paclitaxel on Days 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles or until disease progression whichever occurs first during induction treatment phase. Participants will receive best supportive care during maintenance treatment phase. Switch maintenance to pemetrexed is also permitted. Participants who were consented prior to approval of protocol Version 5 will be given the option to cross over to receive atezolizumab as monotherapy until disease progression.
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin Crossover)
Number analyzed (Participants) | 29 | 20
ng/mL
  Cycle 1 Day 1 Pre-dose: number analyzed (Participants) | 29 | 19
  Cycle 1 Day 1 Pre-dose | NA (NA) — Below the level of detection. | NA (NA) — Below the level of detection.
  Cycle 1 Day 1 Before End of Infusion: number analyzed (Participants) | 23 | 18
  Cycle 1 Day 1 Before End of Infusion | 20,500 (7500) | 17,000 (5200)
  Cycle 1 Day 1 Post Infusion: number analyzed (Participants) | 29 | 18
  Cycle 1 Day 1 Post Infusion | 11,900 (3100) | 12,400 (3800)
  Cycle 3 Day 1 Pre-dose: number analyzed (Participants) | 23 | 16
  Cycle 3 Day 1 Pre-dose | 169 (63.8) | 160 (48.8)
  Cycle 3 Day 1 Before End of Infusion: number analyzed (Participants) | 16 | 14
  Cycle 3 Day 1 Before End of Infusion | 15,300 (6600) | 17,800 (7550)
  Cycle 3 Day 1 Post Infusion: number analyzed (Participants) | 18 | 15
  Cycle 3 Day 1 Post Infusion | 11,400 (3060) | 13,400 (6650)

18. Secondary Outcome: Plasma Concentrations of Nab-Paclitaxel Reported as Total Paclitaxel
Time Frame: Predose (same day of treatment administration), 5-10 minutes before end of nab-paclitaxel infusion, 1 hour after nab-paclitaxel infusion (infusion duration=30 minutes) on Day 1 of Cycle 1 and 3 (1 Cycle=21 days) (up to approximately 35 months)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B (Nab-Paclitaxel+Carboplatin Crossover)
Number analyzed (Participants) | 30 | 20
ng/mL
  Cycle 1 Day 1 Pre-dose: number analyzed (Participants) | 29 | 19
  Cycle 1 Day 1 Pre-dose | NA (NA) — Below the level of detection. | NA (NA) — Below the level of detection.
  Cycle 1 Day 1 Before End of Infusion: number analyzed (Participants) | 27 | 15
  Cycle 1 Day 1 Before End of Infusion | 3520 (2210) | 2530 (1420)
  Cycle 1 Day 1 Post Infusion: number analyzed (Participants) | 25 | 17
  Cycle 1 Day 1 Post Infusion | 307 (153) | 417 (217)
  Cycle 3 Day 1 Pre-dose: number analyzed (Participants) | 23 | 16
  Cycle 3 Day 1 Pre-dose | NA (NA) — Below the threshold of the assay. | NA (NA) — Below the threshold of the assay.
  Cycle 3 Day 1 Before End of Infusion: number analyzed (Participants) | 17 | 10
  Cycle 3 Day 1 Before End of Infusion | 4480 (3520) | 2030 (1690)
  Cycle 3 Day 1 Post Infusion: number analyzed (Participants) | 18 | 15
  Cycle 3 Day 1 Post Infusion | 357 (253) | 447 (322)

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 18 January 2021 (approximately 69 months)
Description: The safety-evaluable population included all treated participants, defined as randomized participants who received any protocol treatment. For the safety analyses, participants were grouped according to whether any full or partial dose of atezolizumab was received, including when atezolizumab was received in error. Specifically, for participants randomized to the CnP arm, if atezolizumab was received in error, the participants were grouped to the Atezo+CnP arm for the safety analyses.
Groups:
- Arm B Without Crossover Participants (Nab-Paclitaxel+Carboplatin): Participants received IV infusion of carboplatin on Day 1 and nab-paclitaxel on Days 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles or until disease progression whichever occurs first during induction treatment phase. Participants received best supportive care during maintenance treatment phase. Switch maintenance to pemetrexed was also permitted. Participants who were consented prior to approval of protocol Version 5 were given the option to cross over to receive atezolizumab as monotherapy until disease progression. This Arm B group includes participants who did not crossover to receive atezolizumab as monotherapy.
- Arm B With Crossover Participants (Nab-Paclitaxel+Carboplatin, After Crossover Atezo Monotherapy): Participants received IV infusion of carboplatin on Day 1 and nab-paclitaxel on Days 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles or until disease progression whichever occurs first during induction treatment phase. Participants received best supportive care during maintenance treatment phase. Switch maintenance to pemetrexed was also permitted. Participants who were consented prior to approval of protocol Version 5 were given the option to cross over to receive atezolizumab as monotherapy until disease progression. This Arm B group includes participants who crossed over to receive atezolizumab as monotherapy.
Arm/Group | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) | Arm B Without Crossover Participants (Nab-Paclitaxel+Carboplatin) | Arm B With Crossover Participants (Nab-Paclitaxel+Carboplatin, After Crossover Atezo Monotherapy)
All-Cause Mortality (participants affected / at risk) | 338/473 | 108/131 | 70/101
Serious Adverse Events (participants affected / at risk) | 252/473 | 63/131 | 24/101
Other Adverse Events (participants affected / at risk) | 467/473 | 127/131 | 100/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) (N=473) | Arm B Without Crossover Participants (Nab-Paclitaxel+Carboplatin) (N=131) | Arm B With Crossover Participants (Nab-Paclitaxel+Carboplatin, After Crossover Atezo Monotherapy) (N=101)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 14 (16) | 4 (4) | 4 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 9 (10) | 3 (3) | 2 (2)
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 14 (16) | 1 (1) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ANEURYSM (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
ADDISON'S DISEASE (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
GLUCOCORTICOID DEFICIENCY (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (5) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 14 (14) | 1 (1) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
GASTROINTESTINAL VASCULAR MALFORMATION HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
IMMUNE-MEDIATED ENTEROCOLITIS (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 3 (4) | 1 (1)
OESOPHAGEAL FOOD IMPACTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 6 (7) | 3 (4) | 1 (1)
ASTHENIA (General disorders) | 3 (5) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 5 (5) | 0 (0) | 0 (0)
DEATH (General disorders) | 1 (1) | 3 (3) | 0 (0)
DRUG INTERACTION (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 1 (1) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 (4) | 1 (1) | 1 (1)
GENERALISED OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (2) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 2 (2) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 3 (3) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN (General disorders) | 2 (2) | 0 (0) | 0 (0)
PERFORMANCE STATUS DECREASED (General disorders) | 2 (2) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 8 (9) | 2 (2) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0) | 0 (0)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
IMMUNE-MEDIATED HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL COLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 6 (6) | 0 (0) | 1 (1)
CAMPYLOBACTER INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
FEBRILE INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
FURUNCLE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GANGRENE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PARAPHARYNGEAL SPACE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 45 (55) | 13 (15) | 2 (2)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 7 (7) | 2 (2) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 6 (6) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 4 (4) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 4 (4) | 2 (3) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
EMBOLIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
TOXIC NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
VASOGENIC CEREBRAL OEDEMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
AUTOIMMUNE NEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
POSTRENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 5 (5) | 1 (1) | 1 (1)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 13 (22) | 5 (8) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (4) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 3 (3) | 2 (2)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
PHLEBITIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
VASCULAR STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Atezolizumab+Nab-Paclitaxel+Carboplatin) (N=473) | Arm B Without Crossover Participants (Nab-Paclitaxel+Carboplatin) (N=131) | Arm B With Crossover Participants (Nab-Paclitaxel+Carboplatin, After Crossover Atezo Monotherapy) (N=101)
ANAEMIA (Blood and lymphatic system disorders) | 259 (357) | 67 (79) | 50 (55)
LEUKOPENIA (Blood and lymphatic system disorders) | 51 (92) | 13 (22) | 6 (7)
NEUTROPENIA (Blood and lymphatic system disorders) | 213 (424) | 52 (95) | 53 (99)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 132 (210) | 29 (49) | 31 (47)
HYPOTHYROIDISM (Endocrine disorders) | 51 (55) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 25 (28) | 2 (2) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 54 (67) | 9 (11) | 8 (9)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 25 (33) | 5 (7) | 6 (7)
CONSTIPATION (Gastrointestinal disorders) | 176 (224) | 38 (47) | 33 (42)
DIARRHOEA (Gastrointestinal disorders) | 196 (321) | 37 (61) | 35 (41)
DRY MOUTH (Gastrointestinal disorders) | 24 (24) | 3 (3) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 33 (34) | 2 (2) | 5 (6)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 24 (25) | 2 (3) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 236 (354) | 61 (85) | 44 (65)
STOMATITIS (Gastrointestinal disorders) | 40 (45) | 8 (9) | 4 (5)
VOMITING (Gastrointestinal disorders) | 130 (228) | 25 (38) | 18 (30)
ASTHENIA (General disorders) | 89 (133) | 19 (26) | 21 (29)
CHEST PAIN (General disorders) | 33 (43) | 10 (10) | 2 (2)
CHILLS (General disorders) | 25 (32) | 4 (4) | 3 (4)
FATIGUE (General disorders) | 228 (297) | 57 (73) | 52 (61)
MUCOSAL INFLAMMATION (General disorders) | 24 (26) | 4 (5) | 4 (4)
OEDEMA PERIPHERAL (General disorders) | 71 (81) | 14 (17) | 11 (13)
PAIN (General disorders) | 30 (33) | 6 (7) | 2 (3)
PYREXIA (General disorders) | 80 (104) | 12 (16) | 10 (15)
BRONCHITIS (Infections and infestations) | 29 (30) | 2 (2) | 4 (5)
NASOPHARYNGITIS (Infections and infestations) | 38 (61) | 4 (4) | 6 (7)
PNEUMONIA (Infections and infestations) | 37 (41) | 6 (6) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 35 (55) | 8 (9) | 4 (6)
URINARY TRACT INFECTION (Infections and infestations) | 63 (91) | 9 (9) | 10 (11)
FALL (Injury, poisoning and procedural complications) | 24 (33) | 4 (4) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 26 (42) | 9 (13) | 5 (5)
BLOOD CREATININE INCREASED (Investigations) | 27 (32) | 7 (11) | 1 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 93 (188) | 18 (33) | 17 (29)
PLATELET COUNT DECREASED (Investigations) | 108 (179) | 22 (29) | 16 (32)
WEIGHT DECREASED (Investigations) | 63 (71) | 15 (16) | 13 (13)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 49 (80) | 9 (16) | 9 (12)
DECREASED APPETITE (Metabolism and nutrition disorders) | 144 (169) | 34 (36) | 30 (34)
DEHYDRATION (Metabolism and nutrition disorders) | 52 (73) | 17 (27) | 8 (8)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 77 (98) | 12 (13) | 12 (16)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 94 (130) | 23 (27) | 17 (23)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 31 (54) | 8 (10) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 113 (161) | 19 (20) | 17 (20)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 89 (105) | 9 (9) | 7 (7)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 25 (27) | 8 (10) | 6 (6)
MYALGIA (Musculoskeletal and connective tissue disorders) | 50 (60) | 5 (5) | 5 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 61 (72) | 7 (7) | 8 (8)
DIZZINESS (Nervous system disorders) | 78 (90) | 14 (21) | 11 (15)
DYSGEUSIA (Nervous system disorders) | 43 (46) | 5 (5) | 7 (7)
HEADACHE (Nervous system disorders) | 85 (106) | 12 (13) | 11 (13)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 56 (58) | 13 (16) | 9 (10)
PARAESTHESIA (Nervous system disorders) | 43 (51) | 7 (7) | 5 (6)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 60 (71) | 10 (14) | 13 (15)
ANXIETY (Psychiatric disorders) | 32 (32) | 4 (4) | 3 (3)
DEPRESSION (Psychiatric disorders) | 29 (29) | 5 (5) | 0 (0)
INSOMNIA (Psychiatric disorders) | 70 (76) | 15 (17) | 16 (16)
COUGH (Respiratory, thoracic and mediastinal disorders) | 135 (162) | 21 (21) | 18 (21)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 134 (181) | 28 (30) | 23 (29)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 69 (84) | 17 (18) | 10 (12)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 30 (42) | 6 (6) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 35 (44) | 4 (4) | 4 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 152 (155) | 33 (33) | 30 (30)
DRY SKIN (Skin and subcutaneous tissue disorders) | 28 (31) | 6 (6) | 6 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 61 (81) | 7 (7) | 5 (5)
RASH (Skin and subcutaneous tissue disorders) | 73 (86) | 6 (7) | 11 (12)
HYPERTENSION (Vascular disorders) | 26 (33) | 3 (4) | 5 (6)
HYPOTENSION (Vascular disorders) | 34 (43) | 6 (8) | 7 (7)
VERTIGO (Ear and labyrinth disorders) | 17 (21) | 2 (2) | 7 (7)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 20 (30) | 8 (10) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 20 (32) | 7 (8) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 20 (21) | 7 (8) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT02367781/Prot_SAP_000.pdf